

# **Clinical Trial Protocol**

| Document Number: | c36231686-05 |
|---|---|
| 2021-004880-28 | |
| 1402-0020 | |
| BI 1358894 | |
| Relative bioavailability of two differ<br>BI 1358894 administered in healthy<br>state (an open-label, randomised, sin<br>sequence crossover study) | subjects in fasted and fed |
| Lay Title A study in healthy people to compare 2 different formulations of BI 1358894 tablets taken with or without food | |
| I | |
| Phone: + , Fax: | + |
| Phone: + Fax: | |
| Version 5.0, 20 Apr 2022 | |
| 11 Oct 2021 | |
| | 2021-004880-28 1402-0020 BI 1358894 Relative bioavailability of two differ BI 1358894 administered in healthy state (an open-label, randomised, sin sequence crossover study) A study in healthy people to compar of BI 1358894 tablets taken with or visible properties. Fax: Phone: + Fax: - Version 5.0, 20 Apr 2022 11 Oct 2021 |

Proprietary confidential information

© 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

# CLINICAL TRIAL PROTOCOL SYNOPSIS

| Company name | Boehringer Ingelheim |
|---|---|
| Original protocol date | 11 Oct 2021 |
| Revision date | 20 Apr 2022 |
| BI trial number | 1402-0020 |
| Title of trial | Relative bioavailability of two different tablet formulations of BI 1358894 administered in healthy subjects in fasted and fed state (an open-label, randomised, single-dose, four-period, four-sequence crossover study) |
| Principal Investigator | |
| Trial site | |
| Clinical phase | I |
| Trial rationale | This trial is conducted to compare the pharmacokinetics of two tablet formulations of BI 1358894 and to assess potential food effects. |
| Trial objective | To investigate the relative bioavailability of the intended Commercial Formulation (iCF) (Test, T) compared with Trial Formulation 2 (TFII) (Reference, R) and to assess potential food effects following oral administration of BI 1358894. |
| Trial endpoints | Primary endpoints: AUC <sub>0-tz</sub> and C <sub>max</sub> of BI 1358894 Secondary endpoints: AUC <sub>0-∞</sub> of BI 1358894 |
| Trial design | Randomised, open-label, single-dose, four-period and four-sequence crossover study |
| Number of subjects | |
| total entered | 24 |
| on each treatment | 24 |
| Diagnosis | Not applicable |
| Main inclusion criteria | Healthy male/female subjects, age of 18 to 55 years (inclusive), body mass index (BMI) of 18.5 to 29.9 kg/m² (inclusive) |
| Test product | BI 1358894, iCF (T), film-coated tablets, dose strength 100 mg |
| dose | 100 mg (1 x 100 mg) |
| mode of<br>administration | Oral administration in fasted (overnight fast of at least 10 hours) and fed state (treatments $T_{\text{fasted}}$ and $T_{\text{fed}}$ ) with 240 mL of water |

c36231686-05 Trial Protocol


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Reference product | BI 1358894, TFII (R), film-coated tablets, dose strength 50 mg |
|---|---|
| dose | 100 mg (2 x 50 mg) |
| mode of admin. | Oral administration in fasted (overnight fast of at least 10 hours) and fed state (treatments $R_{\text{fasted}}$ and $R_{\text{fed}}$ ) with 240 mL of water |
| Duration of treatment | One day (single dose) for each treatment |
| Statistical methods | Relative bioavailability will be estimated by the ratios of the geometric means of the respective pairwise comparison of interest for the primary and secondary endpoints, i.e. for the two tablet formulations under fasted or fed condition and the food effect for each formulation. Additionally, their two-sided 90% confidence intervals (CIs) will be provided. This method corresponds to the two one-sided t-test procedure, each at a 5% significance level. Since the main focus is on estimation and not testing, a formal hypothesis test and associated acceptance range is not specified for any comparison of interest. The statistical model will be an analysis of variance (ANOVA) on the logarithmic scale including effects for sequence, subjects nested within sequences, period and treatment. CIs will be calculated based on the residual error from the ANOVA. Descriptive statistics will be calculated for all endpoints. |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## FLOW CHART

| Period | Visit | Day | Planned time (relative to<br>drug administration)<br>[h:min] | Approximate clock time of actual day [h:min] | Event and comment | Safety laboratory <sup>9</sup> | PK blood | 12-lead ECG | Suicidality Assessessment8 | Vital signs (BP, PR) | Counselling on<br>contraceptive measures <sup>10</sup> | Questioning for AEs and concomitant therapy <sup>6</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SCR | 1 | -21 to -2 | | | Screening (SCR) <sup>1</sup> | xA | | X | X | X | X | |
| | 8 | -1 | -12:00 | 20:00 | Admission to trial site | x <sup>5</sup><br>x <sup>2,B</sup> | | 2 | X | 2 | X | X |
| | | 1 | -1:00 | 07:00 | Allocation to treatment <sup>2</sup> (visit 2 only) | X <sup>2,B</sup> | x <sup>2</sup> | x <sup>2</sup> | | x <sup>2</sup> | | x <sup>2</sup> |
| | | | -0:30 | 07:30 | High fat, high calorie breakfast <sup>7</sup> | | | | | | | |
| | | | 0:00 | 08:00 | Drug administration | | | | | | | |
| bo | | | 0:30 | 08:30 | | | X | | | | | |
| eri | | | 1:00 | 09:00 | | | X | | | | | |
| nt p | | | 1:30 | 09:30 | | | X | | | | | |
| ō | | | 2:00 | 10:00 | 240 mL fluid intake | | X | | | | | |
| ash | | | 3:00 | 11:00 | | | X | | | | | |
| y a w | | | 4:00 | 12:00 | 240 mL fluid intake, thereafter lunch <sup>3</sup> | | X | | | X | | X |
| ods separated by a<br>of at least 17 days | | | 5:00 | 13:00 | | | X | | | | | |
| ate | 2/3/4/5 | | 6:00 | 14:00 | | | X | | | | | |
| par | /3/ | | 7:00 | 15:00 | | | X | | | | | |
| s se | C | | 8:00 | 16:00 | | | X | | | X | | |
| spo<br>of a | | | 10:00 | 18:00 | Dinner <sup>3</sup> | | X | | | | | |
| eri | | | 12:00 | 20:00 | | | X | | | | | X |
| 1/2/3/4 (four periods separated by a wash-out period of at least 17 days | | 2 | 24:00 | 08:00 | Breakfast (voluntary) <sup>3</sup> ,<br>discharge from trial site | xB | X | | | X | X | X |
| 4 ( | | | 34:00 | 18:00 | Ambulatory visit | | X | | | X | | X |
| 2/3/ | | 3 | 48:00 | 08:00 | Ambulatory visit | | X | | | | | X |
| 1/2 | | 4 | 72:00 | 08:00 | Ambulatory visit | | X | | | | | X |
| | | 5 | 96:00 | 08:00 | Ambulatory visit | | X | | | | | X |
| | | 6 | 120:00 | 08:00 | Ambulatory visit | | X | | | | | X |
| | | 7 | 144:00 | 08:00 | Ambulatory visit | | X | | | | | X |
| | | 11 | 240:00 | 08:00 | Ambulatory visit | xB | X | | | | | X |
| | | 14 | 312:00 | 08:00 | Ambulatory visit | | X | | | | | X |
| FU | 6 | 18 to 25 | | | End of study (EoS)<br>examination <sup>4</sup> | x <sup>C</sup> | | X | X | X | X | х |

- 1. Subject must be informed and written informed consent obtained prior to starting any screening procedures. Screening procedures include physical examination, check of vital signs, ECG, safety laboratory (including drug screening and pregnancy test in female subjects), demographics (including determination of body height and weight, smoking status, alcohol history and suicidality assessment), relevant medical history, concomitant therapy and review of inclusion/exclusion criteria. Pharmacogenetic samples will be collected if needed.
- 2. The time is approximate; the procedure is to be performed and completed within the 3 h prior to drug administration.
- 3. If several actions are indicated at the same time, the intake of meals will be the last action.
- 4. At the end of study (synonym for end of trial), the EoS examination includes physical examination, vital signs, ECG, safety laboratory (including pregnancy test in women), recording of AEs, concomitant therapies and suicidality assessment.
- 5. Only urine drug screening and alcohol breath test as well as pregnancy test in women will be done at this time.
- AEs and concomitant therapies will be recorded throughout the trial, but will be specifically asked for at the times indicated in the Flow Chart above.
- 7. Only for T<sub>fed</sub> and R<sub>fed</sub>

**Boehringer Ingelheim** BI Trial No.: 1402-0020

c36231686-05

20 Apr 2022

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 8. Suicidality assessment using the Columbia-Suicidal Severity Rating Scale (C-SSRS): 'Screening/Baseline' version at Visit 1, and 'since last visit' version at visit 2-6.
- 9. Letter A, B and C define different sets of safety laboratory examinations (see Section 5.2.3).
- 10. For female participants of childbearing potential: counselling on adequate contraceptive measures. At Screening, description of adequate contraceptive measures. Explanation of the background why strict adherence to the measures is required.
  - On day -1, questioning whether contraceptive measures were adhered to.

**Trial Protocol** 

On day 2, and on EoT, reminder to adhere to the contraceptive measures.


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# TABLE OF CONTENTS

| TIT | TLE F | PAGE | 1 |
|----------|-------|----------------------------------------------------|----|
| CL | INIC | AL TRIAL PROTOCOL SYNOPSIS | 2 |
| FL | ow o | CHART | 4 |
| | | OF CONTENTS | |
| | | VIATIONS AND DEFINITIONS | |
| АD<br>1. | | RODUCTION | |
| ı. | | | |
| | 1.1 | MEDICAL BACKGROUND DRUG PROFILE | |
| | 1.2 | 1.2.1 BI 1358894 | |
| | | 1.2.1 BI 1558894 | 13 |
| | 1.3 | RATIONALE FOR PERFORMING THE TRIAL | 15 |
| | 1.4 | BENEFIT - RISK ASSESSMENT | |
| | | 1.4.1 Benefits | |
| | | 1.4.2 Risks | 15 |
| | | | 10 |
| 2. | | IAL OBJECTIVES AND ENDPOINTS | |
| | 2.1 | MAIN OBJECTIVES, PRIMARY AND SECONDARY ENDPOINT | |
| | | 2.1.1 Main objectives | |
| | | 2.1.2 Primary endpoints | |
| | | 2.1.5 Secondary endpoint | 19 |
| | - | 2.2.2.2 Safety and tolerability | 20 |
| 3. | DES | SCRIPTION OF DESIGN AND TRIAL POPULATION | 21 |
| | 3.1 | OVERALL TRIAL DESIGN | 21 |
| | 3.2 | DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE O | F |
| | | CONTROL GROUP | |
| | 3.3 | SELECTION OF TRIAL POPULATION | |
| | | 3.3.1 Main diagnosis for trial entry | |
| | | 3.3.2 Inclusion criteria | |
| | | 3.3.3 Exclusion criteria | |
| | | 3.3.4.1 Withdrawal from trial treatment | |

| c36231686-( | )5 1 | ria | l P | ro | toco |
|-------------|------|-----|-----|----|------|
|-------------|------|-----|-----|----|------|


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Replacement of subjects ......27 4. INVESTIGATIONAL TREATMENTS ......28 Identity of the Investigational Medicinal Products ......28 4.1.2 Selection of doses in the trial......28 Method of assigning subjects to treatment groups ......28 4.1.3 4.1.4 Drug assignment and administration of doses for each subject ......29 4.1.5 Blinding and procedures for unblinding ......30 Packaging, labelling, and re-supply .......31 4.1.6 Storage conditions......31 4.1.7 OTHER TREATMENTS, EMERGENCY PROCEDURES. 4.2 RESTRICTIONS ......32 Other treatments and emergency procedures.......32 4.2.1 Restrictions ......32 4.2.2 TREATMENT COMPLIANCE......33 4.3 5. ASSESSMENT OF EFFICACY......34 5.1 5.2 ASSESSMENT OF SAFETY......34 5.2.1 5.2.2 Vital signs......34 5.2.3 Safety laboratory parameters ......34 5.2.4 5.2.5 Other safety parameters......38 5.2.6.1.4 Adverse events of special interest .......40 

| -2/221/0/ 05 | T 1 D 4 |
|--------------|---------------|
| c36231686-05 | Trial Protoco |


| Proprietary | confidential information © 2022 Boehringer Ingelheim Internation | onal GmbH or one or more of its affiliated companies |
|---|---|---|
|---|---|---|

| | | 5.2.6.2.1 AE collection | |
|----|-----|------------------------------------------------------|----|
| | | 5.2.6.2.2 AE reporting to the sponsor and timelines | |
| | | 5.2.6.2.3 Pregnancy | 43 |
| | | 5.2.6.2.4 AE reporting from suicidality assessment | 43 |
| | 5.3 | DRUG CONCENTRATION MEASUREMENTS AND PHARMACOKINETICS | 44 |
| | | 5.3.1 Assessment of pharmacokinetics | |
| | | 5.3.2 Methods of sample collection | |
| | | 5.3.2.1 Blood sampling for pharmacokinetic analysis | |
| | | 5.3.4 Pharmacokinetic - pharmacodynamic relationship | |
| | 5.4 | ASSESSMENT OF BIOMARKERS | |
| | 5.5 | BIOBANKING | |
| | 5.6 | OTHER ASSESSMENTS | |
| | | 5.6.1 Pharmacogenomic evaluation | |
| | 5.7 | APPROPRIATENESS OF MEASUREMENTS | |
| 6. | INV | ESTIGATIONAL PLAN | 47 |
| | 6.1 | VISIT SCHEDULE | 47 |
| | 6.2 | DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS | 47 |
| | | 6.2.1 Screening | 47 |
| | | 6.2.2 Treatment period | |
| | | 6.2.3 Follow-up period and trial completion | 48 |
| 7. | STA | ATISTICAL METHODS AND DETERMINATION OF | |
| | SAN | MPLE SIZE | 49 |
| | 7.1 | NULL AND ALTERNATIVE HYPOTHESES | 49 |
| | 7.2 | PLANNED ANALYSES | 49 |
| | | 7.2.1 General considerations | 49 |
| | | 7.2.1.1 Analysis sets | |
| | | 7.2.1.2 Pharmacokinetics | 50 |
| | | 7.2.2 Primary endpoint analyses | 50 |
| | | 7.2.3 Secondary endpoint analyses | 51 |
| | | 7.2.5 Safety analyses | 52 |
| | | 7.2.6 Interim analyses | |
| | 7.3 | HANDLING OF MISSING DATA | |
| | 7.5 | 7.3.1 Safety | |
| | | 7.3.2 Pharmacokinetics | |
| | 7.4 | RANDOMISATION | |
| | 7.5 | DETERMINATION OF SAMPLE SIZE | |
| | 1.0 | DETERMINATION OF STRIPLE SHEET | |

| 8. | INF | ORMED CONSENT, TRIAL RECORDS, DATA | |
|---|---|---|---|
| | PRC | TECTION, PUBLICATION POLICY, AND | |
| | ADN | MINISTRATIVE STRUCTURE | 56 |
| | 8.1 | TRIAL APPROVAL, SUBJECT INFORMATION, INFORMED | |
| | | CONSENT | |
| | 8.2 | DATA QUALITY ASSURANCE | 57 |
| | 8.3 | RECORDS | 57 |
| | | 8.3.1 Source documents | 57 |
| | | 8.3.2 Direct access to source data and documents | |
| | | 8.3.3 Storage period of records | |
| | 8.4 | EXPEDITED REPORTING OF ADVERSE EVENTS | |
| | 8.5 | STATEMENT OF CONFIDENTIALITY AND SUBJECT PRIVACY | 59 |
| | | 8.5.1 Collection, storage and future use of biological samples and corresponding data | 59 |
| | 8.6 | TRIAL MILESTONES | |
| | 8.7 | ADMINISTRATIVE STRUCTURE OF THE TRIAL | 60 |
| 9. | REF | ERENCES | 62 |
| | 9.1 | PUBLISHED REFERENCES | 62 |
| | 9.2 | UNPUBLISHED REFERENCES | 63 |
| 10. | APP | ENDICES | 65 |
| | 10.1 | COLUMBA-SUICIDE SEVERITY RATING SCALE | 65 |
| 11. | DES | CRIPTION OF GLOBAL AMENDMENTS | 71 |
| | 11.1 | GLOBAL AMENDMENT 1 | 71 |
| | 11.2 | GLOBAL AMENDMENT 2 | 72 |
| | 11.3 | GLOBAL AMENDMENT 3 | 73 |
| | 11.4 | GLOBAL AMENDMENT 4 | 74 |

Boehringer Ingelheim 20 Apr 2022

BI Trial No.: 1402-0020

c36231686-05 Trial Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ABBREVIATIONS AND DEFINITIONS

ADME Absorption, distribution, metabolism, and excretion

AE Adverse event

AESI Adverse events of special interest

ANOVA Analysis of variance

%AUC<sub>tz-∞</sub> Percentage of AUC<sub>0-∞</sub> obtained by extrapolation

AUC<sub>0-tz</sub> Area under the concentration-time curve of the analyte in plasma over the

time interval from 0 to the last quantifiable data point

BA Bioavailability

BI Boehringer Ingelheim

BMI Body mass index (weight divided by height squared)

BP Blood pressure

BPD Borderline personality disorder

CA Competent authority
CI Confidence interval

CL Confidence interval limit

C<sub>max</sub> Maximum measured concentration of the analyte in plasma

CRF Case Report Form, paper or electronic (sometimes referred to as 'eCRF')

C-SSRS Columbia-Suicidal Severity Rating Scale

CT Leader Clinical Trial Leader
CT Manager Clinical Trial Manager
CTP Clinical trial protocol
CTR Clinical trial report
CYP Cytochrome P450

DILI Drug induced liver injury

ECG Electrocardiogram

eCRF Electronic case report form eDC Electronic Data Capture

EDTA Ethylenediaminetetraacetic acid

EoS End of Study (synonym for End of Trial)

EudraCT European Clinical Trials Database

FU Follow-up

GCP Good Clinical Practice

gCV Geometric coefficient of variation HCG Human chorionic gonadotropin Boehringer Ingelheim 20 Apr 2022 BI Trial No.: 1402-0020

c36231686-05 Trial Protocol

White blood cells

WBC

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| $^{\mathrm{IB}}$ | Investigator's brochure |
|---|---|
| iCF | Intended Commercial Formulation |
| IEC | Independent Ethics Committee |
| IPD | Important protocol deviation |
| IRB | Institutional Review Board |
| ISF | Investigator site file |
| MDA | Methylenedioxyamphetamine |
| MDD | Major depressive disorder |
| MDMA | Methylenedioxymethamphetamine |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PK | Pharmacokinetic(s) |
| PKS | Pharmacokinetic parameter analysis set |
| PR | Pulse rate |
| PTSD | Post-traumatic stress disorder |
| qd | Quaque die |
| QT interval | ECG interval from the start of the QRS complex to the end of the T wave |
| QTc interval | QT interval corrected for heart rate, e.g. using the method of Fridericia (QTcF) or Bazett (QTcB) |
| R | Reference treatment |
| REP | Residual effect period |
| SAE | Serious adverse event |
| SCR | Screening |
| SOP | Standard operating procedure |
| T | Test product or treatment |
| TFII | Trial Formulation 2 |
| $t_{max}$ | Time from (last) dosing to the maximum measured concentration of the analyte in plasma |
| TRPC 4/5 | Transient receptor potential cation channel, subfamily C, members 4 and 5 |
| TS | Treated set |
| TSAP | Trial statistical analysis plan |
| $t_z$ | Time of last measurable concentration of the analyte in plasma |
| ULN | Upper limit of normal |


## 1. INTRODUCTION

BI 1358894, an oral, small-molecule inhibitor of a transient receptor potential cation channel, subfamily C, members 4 and 5 (TRPC 4/5) is being developed for major depressive disorder (MDD), borderline personality disorder (BPD), and post-traumatic stress disorder (PTSD).

#### 1.1 MEDICAL BACKGROUND

MDD is a debilitating disease characterized by low mood and often by low self-esteem, low energy, and a loss of interest. It can strongly impact a person's life and health, including significantly increased risk of suicidality, and is difficult to treat, even with systematic antidepressant strategies. In the National Institute of Mental Health funded STAR\*D trial of >4000 patients with nonpsychotic depression, about 30% of the patients did not reach remission after 4 different medications [P06-11895] and continued to experience residual symptoms [R16-5475] that significantly impacted the patients' quality of life [R06-2872]. BPD is a chronic mental disorder with an estimated prevalence of around 2% in the general community [R16-5476] and severely impaired quality of life [R16-5474]. The main symptom clusters of BPD include impulsive-behavioural dyscontrol, cognitive-perceptual symptoms, disturbed interpersonal relations, and affective instability. Patients with BPD have high rates of deliberate self-harm and a rate of completed suicide that is 50 times higher than in the general population [R16-5477]. Even the presence of a single diagnostic feature of BPD is predictive for poor functioning and psychiatric illness burden [R16-5483]. Treatment guidelines recommend psychotherapy as the mainstay of treatment, but pharmacotherapy is commonly used as an adjunctive, symptom-targeted component of treatment. However, no drug is approved for the treatment of BPD.

PTSD is a disabling mental disorder that can develop after first- or second-hand exposure to a traumatic event. Lifetime prevalence in the US was estimated at 6.8%, with 1-year prevalence at 3.6%, but more than twice as high in women (5.2%) than men (1.8%) [R08-4516]. Classic symptoms involve intrusive flashbacks and nightmares of the trauma [R15-4424]. The firstline treatment in adults is psychotherapy, such as cognitive behavioural therapy. Only sertraline and paroxetine (both antidepressants of the serotonin reuptake inhibitor class) have been licensed for the treatment of PTSD in the US, EU, Japan and several other regions globally [R21-1276].



Trial Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1.2 DRUG PROFILE

#### 1.2.1 BI 1358894



c36231686-05

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



## Clinical pharmacology

Overall, 212 healthy volunteers and 25 patients with MDD had been exposed to BI 1358894 in 8 completed Phase I clinical trials.

At the time of CTP writing, 3 Phase I trials in healthy subjects are being analysed and 3 Phase II trials in patients are ongoing.

Single doses of BI 1358894 were administered in the range from 3 mg to 200 mg; Multiple



#### 1.3 RATIONALE FOR PERFORMING THE TRIAL

This trial is conducted to compare the pharmacokinetics of two tablet formulations of BI 1358894 and to assess potential food effects.

#### 1.4 BENEFIT - RISK ASSESSMENT

#### 1.4.1 Benefits

Participation in this clinical trial is without any (therapeutic) benefit for healthy subjects. Their participation, however, is of major importance for the development of BI 1358894.

#### 1.4.2 Risks

Subjects are exposed to risks of trial procedures and risks related to the exposure to the trial medication.

In one completed pivotal embryo-fetal development study in Goettingen minipigs, embryo-fetal development toxicity was identified (decreased number of implantations, increased number of early resorptions, decreased fetal weight, skeletal malformations) at relevant human exposure levels. Maternal toxicity was not seen at human relevant doses. The NOAEL shows that the findings are relevant for the maximum dose (125 mg once daily) tested in the ongoing clinical trials.

Therefore, a risk for teratogenicity in humans cannot be excluded. To mitigate this risk, women of childbearing potential (WOCBP) who are heterosexually active must agree and adhere to contraceptive measures consisting of one highly effective method of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% plus one additional barrier method during the treatment and follow-up period of the trial. Sexual abstinence is also an accepted method for this trial. Pregnancy testing has to be performed at every visit. Additionally, investigators are advised to counsel WOCBP with regard to the importance of contraception at every visit.

c36231686-05 Trial Protocol


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c36231686-05 Trial Protocol


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Risk mitigation SARS-CoV-2 pandemic:

- A risk management plan has been set up at the clinical site that details specific
  precautionary measures (e.g. hygienic rules, wearing of face masks, physical
  distancing), which will be filed in the ISF. These measures were implemented per
  local requirements in Baden-Württemberg and recommendation by the Robert Koch
  Institute. The local requirements may be subject to change and the trial procedures
  will be adapted accordingly, if applicable
- AEs will be closely monitored and guidance pertaining to treatment and management of acute infections occurring during the trial will be provided


c36231686-05 Trial Protocol

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Trial participants will be screened for SARS-CoV-2, e.g. via polymerase chain reaction (PCR) test, prior to screening (see also exclusion criterion 24) and at various time points during the trial
- During the ambulatory visits, subjects are allowed to enter the site only after it was confirmed that subjects do not have any signs or symptoms of infection (e.g. fever)
- In case SARS-CoV-2 infection is suspected in a subject during trial participation, PCR testing will be initiated without delay to enable the investigator to take decisions about the next steps (e.g. according to Section 3.3.4.1)
- Any subject with suspected or diagnosed COVID-19 will be referred to health care professionals in charge to receive treatment according to standard of care



c36231686-05 Trial Protocol


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. TRIAL OBJECTIVES AND ENDPOINTS

## 2.1 MAIN OBJECTIVES, PRIMARY AND SECONDARY ENDPOINTS

## 2.1.1 Main objectives

To investigate the relative bioavailability of the intended Commercial Formulation (iCF) (Test, T) compared with Trial Formulation 2 (TFII) (Reference, R) and to assess potential food effects following oral administration of BI 1358894.

## 2.1.2 Primary endpoints

The following pharmacokinetic parameters will be determined for BI 1358894

- AUC<sub>0-tz</sub> (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)
- C<sub>max</sub> (maximum measured concentration of the analyte in plasma)

## 2.1.3 Secondary endpoint

The following pharmacokinetic parameter will be determined for BI 1358894:

 AUC<sub>0-∞</sub> (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)





## 2.2.2.2 Safety and tolerability

Safety and tolerability of BI 1358894 will be assessed based on:

- Adverse events (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG
- Vital signs (blood pressure, pulse rate)
- Prospective suicidality assessment (C-SSRS)

#### 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

#### 3.1 OVERALL TRIAL DESIGN

The trial will be performed as a randomised, open-label, single-dose, four-period and four-sequence crossover study trial in healthy male and female subjects.

The treatments will be one 100 mg tablet (iCF) of BI 1358894 (test, T) administered to subjects in the fasting ( $T_{fasted}$ ) and fed ( $T_{fed}$ ) state and two 50 mg tablets (TFII) of BI 1358894 (reference, R) administered to subjects in the fasting ( $R_{fasted}$ ) and fed ( $R_{fed}$ ) state. For details, refer to Section 4.1.

The subjects will be randomly allocated to the 4 treatment sequences (see figure 3.1.:1).



Figure 3.1.:1 Trial design

There will be a washout period of at least 17 days between the treatments.

An overview of all relevant trial activities is provided in the <u>Flow Chart</u>. For visit schedule and details of trial procedures at selected visits, refer to Sections 6.1 and 6.2, respectively.

# 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP

For relative bioavailability trials, the crossover design is preferred because of its efficiency: since each subject serves as his/her own control, the comparison between treatments is based on an intra-subject comparison, thus removing inter-subject variability from the comparison between treatments [R94-1529].

c36231686-05


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Also, the washout time of at least 17 days between drug administration of subsequent treatment periods is chosen to diminish the impact of possible carryover effects.

The open-label treatment is not expected to bias results, since the trial endpoints are derived from measurement of plasma concentrations of the analyte, which are provided by a bioanalytical laboratory that is blinded to treatment allocation.

## 3.3 SELECTION OF TRIAL POPULATION

**Trial Protocol** 

It is planned that 24 healthy male and female subjects will enter the trial. They will be recruited from the volunteers' pool of the trial site.

A log of all subjects enrolled into the trial (i.e. who have signed informed consent) will be maintained in the ISF, irrespective of whether they have been treated with investigational drug or not.

## 3.3.1 Main diagnosis for trial entry

The trial will be performed in healthy subjects.

Please refer to Section <u>8.3.1</u> (Source Documents) for the documentation requirements pertaining to the in- and exclusion criteria.

#### 3.3.2 Inclusion criteria

Subjects will only be included in the trial if they meet the following criteria:

- Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12lead ECG, and clinical laboratory tests
- 2. Age of 18 to 55 years (inclusive)
- 3. BMI of 18.5 to 29.9 kg/m<sup>2</sup> (inclusive)
- 4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
- 5. Either male subject, or female subject who meet any of the following criteria for a highly effective contraception from at least 30 days before administration of trial medication until 30 days after trial completion:



**c36231686-05** Trial Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3.3.3 Exclusion criteria

Subjects will not be allowed to participate, if any of the following general criteria apply:

- 1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
- 2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
- 3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
- 4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
- Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
- 6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
- 7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
- 8. History of relevant orthostatic hypotension, fainting spells, or blackouts
- 9. Relevant chronic or acute infections
- 10. Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin
- 11. History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)

- 12. Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
- 13. Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
- 14. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
- 15. Inability to refrain from smoking on specified trial days
- 16. Alcohol abuse (consumption of more than 12 g per day for females and 24 g per day for males)
- 17. Drug abuse or positive drug screening
- 18. Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
- 19. Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
- 20. Inability to comply with the dietary regimen of the trial site
- 21. A marked prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
- 22. A history of additional risk factors for *Torsade de Pointes* (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
- 23. Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
- 24. During COVID-19 pandemic: laboratory test indicative of an ongoing SARS-CoV-2 infection
- 25. For female subjects: Lactation, pregnancy, or plans to become pregnant during the trial or within 30 days after trial completion
- 26. For female subjects: Positive pregnancy test

In addition, the following trial-specific exclusion criteria apply:

- 27. A history of cerebral seizure
- 28. A history of bipolar mood disorder, bulimia or anorexia
- 29. Any lifetime history of suicidal behaviour (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
- 30. Any suicidal ideation of type 2 to 5 on the C-SSRS in the past 12 months (i.e. active suicidal thought, active suicidal thought with method, active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For restrictions of the trial, refer to Section 4.2.2.

## 3.3.4 Withdrawal of subjects from treatment or assessments

Subjects may withdraw or may be removed from trial treatment or may withdraw consent to trial participation as a whole ('withdrawal of consent') with very different implications; please see Sections 3.3.4.1 and 3.3.4.2 below.

If a subject is removed from or withdraws from the trial prior to the first administration of trial medication, the data of this subject will not be entered in the case report form (CRF) and will not be reported in the clinical trial report (CTR).

If a subject is removed from or withdraws from the trial after the first administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF; in addition, trial data will be included in the CRF and will be reported in the CTR.

Following removal or withdrawal, a complete end-of-trial examination should be performed. If the discontinuation or withdrawal occurs before the end of the REP (see Section 1.2.2, the discontinued subject should, if possible, be questioned for AEs and concomitant therapies at or after the end of the REP, in order to ensure collection of AEs and concomitant therapies throughout the REP, if not contrary to any consent withdrawal of the subject.

#### 3.3.4.1 Withdrawal from trial treatment

An individual subject will be withdrawn from trial treatment if:

- 1. The subject wants to withdraw from trial treatment. The subject will be asked to explain the reasons but has the right to refuse to answer
- 2. The subject has repeatedly shown to be non-compliant with important trial procedures and, in the opinion of both, the investigator and sponsor representative, the safety of the subject cannot be guaranteed as he / she is not willing or able to adhere to the trial requirements in the future.
- 3. The subject needs to take concomitant medication that interferes with the investigational medicinal product or other trial treatment
- 4. The subject can no longer receive trial treatment for medical reasons (such as pregnancy, surgery, adverse events (AEs), or diseases). Specifically the subject will not receive further trial treatment if he/she experiences a severe adverse drug reaction (i.e. a severe adverse event judged to be related to trial medication).
- 5. The subject has an elevation of AST and/or ALT ≥3-fold ULN <u>and</u> an elevation of total bilirubin ≥2-fold ULN (measured in the same blood sample) and/or needs to be followed up according to the DILI checklist provided in the electronic data capture (EDC) system.
- 6. The subject exhibits serious suicidality, in the clinical judgment of the investigator or according to the following criteria:
  - Any suicidal behaviour (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)

• Any suicidal ideation of type 2, 3, 4 or 5 in the C-SSRS (i.e. active suicidal thought without method, intent or plan; active suicidal thought with method but without intent or plan; active suicidal thought with method and intent but without specific plan; or active suicidal thought with method, plan and intent)

In addition to these criteria, the investigator may discontinue subjects at any time based on his or her clinical judgment.

If it is known that a subject becomes pregnant during the trial, administration of the trial medication is to be stopped immediately, and the subject is to be removed from the trial. The subject is to be followed until she has given birth or until the end of the pregnancy. The subject's data are to be collected until the end of the trial (last visit of last subject) and reported in the CTR. For reporting of pregnancy and associated events, refer to Section 5.2.6.2.3.

If new efficacy or safety information becomes available, Boehringer Ingelheim will review the benefit-risk-assessment and, if needed, pause or discontinue the trial treatment for all subjects or take any other appropriate action to guarantee the safety of the trial subjects.

## 3.3.4.2 Withdrawal of consent to trial participation

Subjects may withdraw their consent to trial participation at any time without the need to justify the decision. If a subject wants to withdraw consent, the investigator should be involved in the discussion with the subject and explain the difference between trial treatment discontinuation and withdrawal of consent to trial participation, as well as explain the options for continued follow-up after trial treatment discontinuation, please see Section 3.3.4.1 above.

## 3.3.4.3 Discontinuation of the trial by the sponsor

Boehringer Ingelheim reserves the right to discontinue the trial at any time for any of the following reasons (if reasons 4 and/or 5 are met, the trial should be discontinued immediately):

- 1. Failure to meet expected enrolment goals overall or at a particular trial site
- The sponsor decides to discontinue the further development of the investigational products
- 3. Deviation from GCP, or the CTP impairing the appropriate conduct of the trial
- 4. New toxicological findings, serious adverse events, or any safety information invalidating the earlier positive benefit-risk-assessment (see Section 3.3.4.1)
- More than 50% of the subjects show drug-related and clinically relevant adverse events of moderate or severe intensity, or if at least one drug-related serious adverse event is reported

The trial will be at least temporarily halted if two or more severe adverse reactions (i.e. severe adverse events judged to be related to trial medication) are reported.

Boehringer Ingelheim BI Trial No.: 1402-0020

c36231686-05 Trial Protocol

20 Apr 2022


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3.3.5 Replacement of subjects

In case more than 4 subjects do not complete the trial (including subjects non- evaluable for PK), subjects may be replaced if considered necessary to reach the objective of the trial. Subjects who withdraw or are withdrawn from treatment or assessments because of a drug-related adverse event will not be replaced. The Clinical Trial Leader together with the Trial Pharmacokineticist and the Trial Statistician are to decide, if and how many subjects will be replaced. The total number of replacements may not exceed 1/3 of the total number of evaluable subjects anticipated to complete the trial. A replacement subject will be assigned a unique trial subject number, and will be assigned to the same treatment sequence as the subject he or she replaces.

Boehringer Ingelheim 20 Apr 2022

BI Trial No.: 1402-0020

c36231686-05 Trial Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4. TREATMENTS

#### 4.1 INVESTIGATIONAL TREATMENTS

## 4.1.1 Identity of the Investigational Medicinal Products

The characteristics of the test product (T) are given below:

Substance: BI 1358894

Pharmaceutical formulation: film-coated tablet, iCF

Source: BI Pharma GmbH & Co. KG, Germany

Unit strength: 100 mg
Posology: 1-0-0
Mode of administration: Oral

The characteristics of the reference product (R) are given below:

Substance: BI 1358894

Pharmaceutical formulation: film-coated tablet, TFII (conventional form: C1)

Source: BI Pharma GmbH & Co. KG, Germany

Unit strength: 50 mg
Posology: 2-0-0
Mode of administration: Oral

#### 4.1.2 Selection of doses in the trial

The dose selected for this trial is one of the standard clinical doses (see Section 1.2).

## 4.1.3 Method of assigning subjects to treatment groups

The randomisation scheme will be provided to the trial site in advance. Subjects will be allocated to treatment sequences prior to the first administration of trial medication in the morning of Day 1 (Visit 2). For this purpose, numbers of the randomisation

c36231686-05

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

scheme will be allocated to the subjects by drawing lots. Subjects are then assigned to a treatment sequence according to the randomisation scheme. Once a subject number has been assigned, it cannot be reassigned to any other subject. All subjects may be treated in one cohort, i.e. all subjects may receive treatment on the same calendar day. In case this is not feasible (e.g., due to logistical or recruitment reasons), the group may be split into several cohorts as required. Treatment of all subjects on the same calendar day is acceptable based on the data available for BI 1358894. For discussion of trial-associated risks and safety measures, see Section 1.4).

The randomisation procedure is described in Section 7.4.

**Trial Protocol** 

#### 4.1.4 Drug assignment and administration of doses for each subject

This is a 4-way crossover trial. All subjects will receive the 4 treatments in randomised order. The treatments to be evaluated are summarised in Table 4.1.4: 1 below.

Table 4.1.4: 1 Dosage and treatment schedule

| Treatment | Substance | Formulation | Unit strength | Dosage | Metabolic state | Total dose |
|---|---|---|---|---|---|---|
| $T_{fasted}$ | BI 1358894 | iCF | 100 mg | 1 film-coated tablet qd | Fasted | 100 mg |
| $T_{\tt fed}$ | BI 1358894 | iCF | 100 mg | 1 film-coated tablet qd | Fed | 100 mg |
| $R_{\text{fasted}}$ | BI 1358894 | TFII | 50 mg | 2 film-coated tablets qd | Fasted | 100 mg |
| $R_{\text{fed}}$ | BI 1358894 | TFII | 50 mg | 2 film-coated tablets qd | Fed | 100 mg |

Administration of trial medication in two treatment periods (treatments T<sub>fasted</sub> and R<sub>fasted</sub>) will be performed after subjects have fasted overnight; fasting is to start no later than 10 h before the scheduled dosing. The investigator (or authorised designee) will administer the trial medication as an oral dose together with about 240 mL of water to subjects who are in a standing position. For drug administration, the so-called four-eye principle (two-person rule) should be applied. For this, one authorised employee of the trial site should witness the administration of trial medication, and – if applicable – its preparation, if correct dosage cannot be ensured otherwise. In two treatment periods (treatments T<sub>fed</sub> and R<sub>fed</sub>), the subjects will start to consume a high-fat, high-calorie meal 30 min before drug administration. The subjects must completely consume the meal prior to drug intake. The composition of the standard high-fat, high-calorie meal is detailed in Table 4.1.4: 2; this meal is in compliance with the FDA guidance 'Food-Effect Bioavailability and Fed Bioequivalence Studies' [RO3-2269]. For restrictions with regard to diet, see Section 4.2.2.2.


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 4.1.4: 2 Composition of the high-fat, high-calorie meal

| Ingredients | kcal |
|---------------------------------------------------|------|
| 2 chicken eggs (whole content) for scrambled eggs | 192 |
| 10 g butter for frying scrambled eggs | 75 |
| 35 g fried bacon | 186 |
| 2 toasted slices of wheat bread | 130 |
| 15 g butter for buttering toast slices | 113 |
| 115 g hash brown potatoes | 132 |
| 240 mL whole milk (3.5% fat) | 156 |
| Sum <sup>1</sup> | 984 |

The total caloric content was supplied approximately as following: 150 kcal as protein, 250 kcal as carbohydrate, and 500 to 600 kcal as fat.

Subjects will be kept under close medical surveillance until 24 h after drug administration. During the first 4 h after drug administration, subjects are not allowed to lie down (i.e. no declination of the upper body of more than 45 degrees from upright posture).

The treatments will be separated by a wash-out phase of at least 17 days.

## 4.1.5 Blinding and procedures for unblinding

The table below summarizes the masking/blinding level of individual functions, roles and responsibilities involved in the trial.

Table 4.1.5: 1 Blinding level of individual functions

| Role/function | Timing of receiving access to the treatment information (including rationale) |
|---|---|
| Subject/Participant | This open label trial will provide the subject treatment information as soon as treatment has been assigned. |
| Investigator/Site Staff | The randomization scheme will be provided to the trial site prior to first subject entered for preparation of medication. |
| Sponsor trial team and data | Unblinded as requested. |
| Bioanalytical Staff | Persons directly involved in bioanalyses of PK samples will be blinded to trial treatments. |
| Pharmacokineticist/<br>Pharmacometrician | As requested for analysis. |
| Unblinded Pharmacist/<br>Pharmacy staff | Prior to first subject entered. |

During the time a role/function is blinded according to the table above, the randomisation schemes (i.e. the treatment information) are kept restricted by the global Randomization Team per Sponsor SOP.

PK samples will be labelled in such a way that treatment allocation cannot be derived by the analytical site.

## 4.1.6 Packaging, labelling, and re-supply

The investigational medicinal products will be provided by BI. They will be packaged and labelled in accordance with the principles of Good Manufacturing Practice (GMP).

For details of packing and the description of the label, refer to the ISF.

The telephone number of the sponsor and the name address and telephone number of the trial site are provided in the subject information form. The EudraCT number is indicated on the title page of this protocol as well as on the subject information and informed consent forms.

Packaging and labelling will be performed in such a way that reserve samples as per 21CFR320 are available for storage by the investigational site and that the trial materials can be chosen in a random way by the Investigator.

No re-supply is planned.

## 4.1.7 Storage conditions

Drug supplies will be kept in their original packaging and in a secure limited access storage area in accordance with the recommended (labelled) storage conditions. If necessary, a temperature log must be maintained to make certain that the drug supplies are stored at the correct temperature. If the storage conditions are found to be outside the specified range, the Clinical Research Associate (as provided in the list of contacts) is to be contacted immediately.

## 4.1.8 Drug accountability

The investigator or designee will receive the investigational drugs delivered from the sponsor when the following requirements are fulfilled:

- Approval of the clinical trial protocol by the IRB / ethics committee
- Approval/notification of the regulatory authority, e.g. competent authority
- Availability of the *curriculum vitae* of the Principal Investigator
- Availability of a signed and dated clinical trial protocol

Only authorised personnel documented in the form 'Trial Staff List' may dispense investigational drugs to trial subjects. Investigational drugs are not allowed to be used outside of this protocol.

The investigator or designee must maintain records of the product's delivery to the trial site, the inventory at the site, the use by each subject, and the disposal of unused products. These records will include dates, quantities, batch / serial numbers, expiry ('use-by') dates, and the unique code numbers assigned to the investigational medicinal product and trial subjects.

c36231686-05

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The investigator or designee will maintain records that document adequately that the subjects were provided the doses specified by the CTP and reconcile all investigational medicinal products received from the sponsor. At the time of disposal of remaining trial medication, the investigator or designee must verify that no remaining supplies are in the investigator's possession.

All unused medication will be disposed of locally by the trial site upon written authorisation of the Clinical Trial Leader. Receipt, usage and disposal of trial medication must be documented on the appropriate forms. Account must be given for any discrepancies.

# 4.2 OTHER TREATMENTS, EMERGENCY PROCEDURES, RESTRICTIONS

## 4.2.1 Other treatments and emergency procedures

**Trial Protocol** 

There are no special emergency procedures to be followed. No additional treatment is planned. However, if adverse events require treatment, the investigator can authorise symptomatic therapy. In those cases, subjects will be treated as necessary and, if required, kept under supervision at the trial site or transferred to a hospital until all results of medical evaluations are acceptable.

#### 4.2.2 Restrictions

## 4.2.2.1 Restrictions regarding concomitant treatment

In principle, no concomitant therapy is allowed except for hormonal contraceptives, hormonal replacement therapy, and SARS-CoV2 vaccination. All concomitant or rescue therapies will be recorded (including time of intake on trial days) on the appropriate pages of the CRF.

## 4.2.2.2 Restrictions on diet and life style

While admitted to the trial site, the subjects will be instructed not to consume any foods or drinks other than those provided by the staff. Standardised meals will be served at the times indicated in the <u>Flow Chart</u>. No food is allowed for at least 4 h after drug intake.

From 1 h before drug intake until lunch, fluid intake is restricted to the milk served with breakfast (see Table 4.1.4: 2), the water administered with the drug, and an additional 240 mL of water at 2 h and 4 h post-dose (mandatory for all subjects). From lunch until 24 h post-dose, total fluid intake is restricted to 3000 mL.

Alcoholic beverages, grapefruits, Seville oranges (sour or bitter oranges) and their juices, and dietary supplements and products containing St. John's wort (*Hypericum perforatum*) are not permitted from 7 days before the first administration of trial medication until after the last PK sample of each trial period is collected.

Poppy-seeds containing foods should not be consumed within 3 days before each admission to trial site, in order to avoid false-positive results in the drug screen.

c36231686-05 Trial Protocol

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Methylxanthine-containing drinks or foods (such as coffee, tea, cola, energy drinks, or chocolate) are not allowed from 24 h before until 24 h after each administration of trial medication.

Smoking is not allowed during in-house confinement.

Excessive physical activity (such as competitive sport) should be avoided from 7 days before the first administration of trial medication until the end of trial examination.

Direct exposure to the sun or exposure to solarium radiation should be avoided during the entire trial.

## 4.2.2.3 Contraception requirements

If female subjects of child-bearing potential are included in the trial, adequate contraception is to be maintained throughout the course of the trial (see Section 3.3.2 for the definition of adequate measures).

#### 4.3 TREATMENT COMPLIANCE

Compliance will be assured by administration of all trial medication in the trial centre under supervision of the investigating physician or a designee. The measured plasma concentrations of trial medication will provide additional confirmation of compliance.

Subjects who are non-compliant (for instance, who do not appear for scheduled visits or violate trial restrictions) may be removed from the trial and the CRF will be completed accordingly (for further procedures, please see Section 3.3.4.1).


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5. ASSESSMENTS

#### 5.1 ASSESSMENT OF EFFICACY

Not applicable.

## 5.2 ASSESSMENT OF SAFETY

#### 5.2.1 Medical examination

At screening, the medical examination will include demographics, height and body weight, smoking and alcohol history (alcohol history not mandatory to be entered into CRF or to be reported), relevant medical history and concomitant therapy, review of inclusion and exclusion criteria, review of vital signs (BP, PR), 12-lead ECG, laboratory tests, and a physical examination. At the end of trial examination, it will include review of vital signs, 12-lead ECG, laboratory tests, and a physical examination.

Suicidality assessment (see section 5.2.5.1) is performed at the timepoints indicated in the Flow Chart.

## 5.2.2 Vital signs

Systolic and diastolic blood pressures (BP) as well as pulse rate (PR) or heart rate (heart rate is considered to be equal to pulse rate) will be measured by a blood pressure monitor (Dinamap Pro 100, at the times indicated in the Flow Chart, after subjects have rested for at least 5 min in a supine position. All recordings should be made using the same type of blood pressure recording instrument on the same arm, if possible.

## 5.2.3 Safety laboratory parameters

For the assessment of laboratory parameters, blood and urine samples will be collected by the trial site at the times indicated in the Flow Chart after the subjects have fasted for at least 9 h. For retests, at the discretion of the investigator or designee, overnight fasting is not required.

The parameters to be assessed are listed in Tables <u>5.2.3: 1</u> and <u>5.2.3: 2</u>. Reference ranges will be provided in the ISF.

Manual differential white blood cell count or urine sediment examinations will only be performed if there is an abnormality in the automatic blood cell count or in the urinalysis, respectively.


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 5.2.3: 1 Routine laboratory tests

| Functional lab group | BI test name [comment/abbreviation] | A | В | C |
|---|---|---|---|---|
| Haematology | Haematocrit | X | X | X |
| in a superference on the second | Haemoglobin | X | X | X |
| | Red Blood Cell Count/Erythrocytes | | X | X |
| | White Blood Cells/Leucocytes | | X | X |
| | Platelet Count/Thrombocytes (quant) X | | $\mathbf{X}$ | X |
| | Erythrocyte Sedimentation Rate 1 h | X | X | X |
| Automatic WBC | Neutrophils/Leukocytes; Eosinophils/Leukocytes; Basophils/ | X | X | X |
| differential, relative | Leukocytes; Monocytes/Leukocytes; | approximate and approximate an | | |
| Mayoria Control of Anna Contro | Lymphocytes/Leukocytes | | | |
| Manual differential | Neut. Poly (segs)/Leukocytes; Neutrophils | | | |
| WBC (if automatic | Bands/Leukocytes; Eosinophils/Leukocytes; | | | |
| differential WBC is | Basophils/ Leukocytes; | | | |
| abnormal) | Monocytes/Leukocytes; | | | |
| | Lymphocytes/Leukocytes | | | |
| Coagulation | Activated Partial Thromboplastin Time | X | 222 | 22 |
| | Prothrombin time | X | 2027 | 22 |
| | Prothrombin time – INR (International Normalization Ratio) | X | == | |
| Enzymes | AST [Aspartate aminotransferase] /GOT, SGOT | X | X | X |
| | ALT [Alanine aminotransferase] /GPT, SGPT | X | X | X |
| | Alkaline Phosphatase | X | X | X |
| | Gamma-Glutamyl Transferase | X | X | X |
| | Creatine Kinase [CK] | X | 222 | 20 |
| | Creatine Kinase Isoenzyme MB [only if CK is elevated] | X | 222 | 22 |
| Hormones | Thyroid Stimulating Hormone | X | | |

| Substrates | Glucose (Plasma) | X | X | X | ſ |
|------------|----------------------------|---|---|---|---|
| | Creatinine | X | X | X | ı |
| | GFR/ CKD-EPI | X | X | X | ı |
| | Bilirubin, Total | X | X | X | ı |
| | Bilirubin, Direct | X | X | X | ı |
| | Protein, Total | X | X | X | ı |
| | C-Reactive Protein (Quant) | X | X | X | |

<sup>\*</sup> In male subjects only


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 5.2.3: 1 Routine laboratory tests (cont.)

| Functional lab group | BI test name [comment/abbreviation] | A | В | C |
|---|---|---|---|---|
| Electrolytes | Sodium | X | X | X |
| | Potassium | X | $\mathbf{X}$ | X |
| Urinalysis (Stix) | Urine Nitrite (qual) | X | | X |
| 20 20 00 | Urine Protein (qual) | X | | X |
| | Urine Glucose (qual) | X | == | X |
| | Urine Ketone (qual) | X | | X |
| | Urobilinogen (qual) | $\mathbf{X}$ | | X |
| | Urine Bilirubin (qual) | X | | X |
| | Urine RBC/Erythrocytes (qual) | $\mathbf{X}$ | | X |
| | Urine WBC/Leucocytes (qual) | X | | X |
| | Urine pH | X | | X |
| Urine sediment | Only positive findings will be reported (for instance, the | | | |
| (microscopic | presence of sediment bacteria, casts in sediment, squamous | | | |
| examination if | epithelial cells, erythrocytes, leukocytes) | | | |
| erythrocytes, | | | | |
| leukocytes nitrite or | | | | |
| protein are abnormal in | | | | |
| urine) | | | | |

A: parameters to be determined at Visit 1 (screening examination)

The tests listed in Table <u>5.2.3: 2</u> are exclusionary laboratory tests that may be repeated as required. The results will not be entered in the CRF/database and will not be reported in the CTR. Except for pregnancy tests and drug screening, it is planned to perform these tests during screening only. Pregnancy testing in women will be performed at screening, prior to each treatment period, and as part of the end of trial examination. Drug screening will be performed at screening and prior to each treatment period.

B: parameters to be determined at Visit 2, 3, 4 and 5 (for time points refer to Flow Chart)

C: parameters to be determined at Visit 6 (end of trial examination)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 5.2.3: 2 Exclusionary laboratory tests

| Functional lab group | Test name |
|---|---|
| Drug screening (urine) | Amphetamine/MDA Barbiturates Benzodiazepine Cannabis |
| | Cocaine Methadone Methamphetamines/MDMA/Ecstasy Opiates Phencyclidine Tricyclic antidepressants |
| Infectious serology (blood) | Hepatitis B surface antigen (qualitative) Hepatitis B core antibody (qualitative) Hepatitis C antibodies (qualitative) HIV-1 and HIV-2 antibody (qualitative) |
| Pregnancy test (urine) | Beta human chorionic gonadotropin (beta-HCG) |

To encourage compliance with alcohol restrictions, a breath alcohol test (e.g. AlcoTrue® M, will be performed prior to each treatment period, and may be repeated at any time during the trial at the discretion of an investigator or designee. The results will not be included in the CTR.

The laboratory tests listed in Tables 5.2.3: 1 and 5.2.3: 2 will be performed at , with the exception of drug screening and pregnancy tests. These tests will be performed at the trial site using M-10/14-PDT Surestep Multiline test and HCG-K20 test, respectively, or comparable test systems.

Laboratory data will be transmitted electronically from the laboratory to the trial site.

It is the responsibility of the Investigator to evaluate the laboratory reports. Clinically relevant abnormal findings as judged by the Investigator are to be reported as adverse events (please refer to Section 5.2.6).

In case the criteria for hepatic injury are fulfilled, a number of additional measures will be performed (please see Section 5.2.6.1.4).

#### 5.2.4 Electrocardiogram



To achieve a stable heart rate at rest and to assure high quality recordings, the site personnel will be instructed to assure a relaxed and quiet environment, so that all subjects are at complete rest.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

All ECGs will be recorded for a 10 sec duration after subjects have rested for at least 5 min in a supine position. ECG assessment will always precede all other trial procedures scheduled for the same time to avoid compromising ECG quality.

All ECGs will be stored electronically on the Muse CV Cardiology System (
). Electrode placement will be performed according to the method of Wilson, Goldberger and Einthoven.

All locally printed ECGs will be evaluated by the investigator or a designee. Abnormal findings will be reported as AEs (during the trial) or baseline conditions (if identified at the screening visit) if assessed to be clinically relevant by the investigator. Any ECG abnormalities will be carefully monitored and, if necessary, the subject will be removed from the trial and will receive the appropriate medical treatment.

ECGs may be repeated for quality reasons (for instance, due to alternating current artefacts, muscle movements, or electrode dislocation) and the repeated ECG will be used for analysis. Additional (unscheduled) ECGs may be collected by the investigator for safety reasons.

#### 5.2.5 Other safety parameters

#### 5.2.5.1 Suicidality assessment

The C-SSRS is a semi-structured, investigator-rated interview, developed by clinical experts in cooperation with the FDA, assessing both suicidal behaviour and suicidal ideation. It does not give a global score, but provides some categorical and some severity information specifically for behaviour and ideation [R08-1147].

The C-SSRS interview may be administered by any type of physician, psychologist, clinical social worker, mental health counsellor, nurse, or coordinator with C-SSRS training. It has a typical duration of five minutes, and causes only a low burden on subjects. At a minimum, the interview consists of 2 screening questions related to suicidal ideation and 4 related to suicidal behaviour, and may be expanded to up to 17 items in case of positive responses. Free text entries are allowed.

The C-SSRS has been widely used in large multinational CTs. The C-SSRS will be administered at the screening visit (using the 'screening / baseline' version) with the aim to exclude subjects with active moderate or severe symptomatology within a specified time prior to the screening or baseline visit. The life time history of suicidal ideation and behaviour will also be recorded. See Section 10.1 for the original English C-SSRS. For this trial, the paper version of the respective German translation will be used. After the screening visit, the 'since last visit' version is used for the suicidality assessment at the time points indicated in the Flow Chart.

Positive reports are generated for any of the following findings:

Suicidal ideation

- Suicidal ideation with intention to act (type 4)
- Suicidal ideation with specific plan and intent (type 5)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Suicidal behaviour

c36231686-05

- Completed suicide
- Suicide attempt
- Interrupted attempt
- Aborted attempt
- Preparatory actions toward imminent suicidal behaviours.

**Trial Protocol** 

**Negative** reports of suicidal ideation are defined as reports when there are no indications of the above, i.e. suicidal ideation of type 1-3.

The investigator is to review positive and negative reports for plausibility and clinical relevance. Doubtful reports may be repeated or reports may be validated by a consulting psychiatrist.

If there is a confirmed positive report of suicidal behaviour or suicidal ideation type 4 or 5 after start of trial, the investigator is to immediately interview the subject during the clinic visit, and/or is to consult a psychiatrist. If the positive report is confirmed, appropriate actions for the subject's safety have to be initiated.

For details regarding AE reporting see section <u>5.2.6.2.4</u>

#### 5.2.6 Assessment of adverse events

#### 5.2.6.1 Definitions of adverse events

#### 5.2.6.1.1 Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether considered related or not.

The following should also be recorded as an AE in the CRF and BI SAE form (if applicable):

- Worsening of the underlying disease or of other pre-existing conditions
- Changes in vital signs, ECG, physical examination, and laboratory test results, if they
  are judged clinically relevant by the investigator

If such abnormalities already pre-exist prior to trial inclusion, they will be considered as baseline conditions and should be collected in the eCRF only.

#### 5.2.6.1.2 Serious adverse event

A serious adverse event (SAE) is defined as any AE which fulfils at least one of the following criteria:

- Results in death
- Is life-threatening, which refers to an event in which the patient was at risk of death
  at the time of the event; it does not refer to an event that hypothetically might have
  caused death if more severe
- Requires inpatient hospitalisation, or prolongation of existing hospitalisation
- Results in persistent or significant disability or incapacity
- Is a congenital anomaly/birth defect
- Is deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgment which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of dependency or abuse

#### 5.2.6.1.3 AEs considered 'Always Serious'

In accordance with the European Medicines Agency initiative on Important Medical Events, Boehringer Ingelheim has set up a list of AEs, which, by their nature, can always be considered to be 'serious' even though they may not have met the criteria of an SAE as defined above.

The latest list of 'Always Serious AEs' can be found in the eDC system, an electronic data capture system which allows the entry of trial data at the trial site. A copy of the latest list of 'Always Serious AEs' will be provided upon request. These events should always be reported as SAEs as described in Section 5.2.6.2.

Cancers of new histology must be classified as a serious event regardless of the time since discontinuation of the trial medication and must be reported as described in 5.2.6.2, subsections 'AE Collection' and 'AE reporting to sponsor and timelines'.

#### 5.2.6.1.4 Adverse events of special interest

The term adverse events of special interest (AESI) relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class. AESIs need to be reported to the sponsor's Pharmacovigilance Department within the same timeframe that applies to SAEs, please see Section 5.2.6.2.2.

BI Trial No.: 1402-0020

C36231686-05 Trial Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The following are considered as AESIs:

#### Potential severe DILI

A potential severe Drug Induced Liver Injury (DILI) that requires follow-up is defined by the following alterations of hepatic laboratory parameters:

- o An elevation of AST (aspartate aminotransferase) and/or ALT (alanine aminotransferase) ≥3-fold ULN combined with an elevation of total bilirubin ≥2-fold ULN measured in the same blood sample, or in samples drawn within 30 days of each other, or
- o Aminotransferase (ALT, and/or AST) elevations ≥10-fold ULN

These lab findings constitute a hepatic injury alert and the subjects showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided via eDC. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure that these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

#### 5.2.6.1.5 Intensity (severity) of AEs

The intensity (severity) of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) that is/are easily tolerated Moderate: Sufficient discomfort to cause interference with usual activity

Severe: Incapacitating or causing inability to work or to perform usual activities

#### 5.2.6.1.6 Causal relationship of AEs

Medical judgment should be used to determine whether there is a reasonable possibility of a causal relationship between the AE and the given trial treatment, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest that there is a reasonable possibility of a causal relationship could be:

- The event is consistent with the known pharmacology of the drug
- The event is known to be caused by or attributed to the drug class
- A plausible time to onset of the event relative to the time of drug exposure
- Evidence that the event is reproducible when the drug is re-introduced
- No medically sound alternative aetiologies that could explain the event (e.g. preexisting or concomitant diseases, or co-medications)
- The event is typically drug-related and infrequent in the general population not exposed to drugs (e.g. Stevens-Johnson syndrome)

• An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is reduced)

Arguments that may suggest that there is no reasonable possibility of a causal relationship could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days / weeks of drug administration; an allergic reaction weeks after discontinuation of the drug concerned)
- Continuation of the event despite the withdrawal of the medication, taking into account the pharmacological properties of the compound (e.g. after 5 half-lives). Of note, this criterion may not be applicable to events whose time course is prolonged despite removing the original trigger
- There is an alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned
- Disappearance of the event even though the trial drug treatment continues or remains unchanged
- 5.2.6.2 Adverse event collection and reporting

#### 5.2.6.2.1 AE collection

Upon enrolment into a trial, the subject's baseline condition is assessed (for instance, by documentation of medical history/concomitant diagnoses), and relevant changes from baseline are noted subsequently.

Subjects will be required to report spontaneously any AEs. In addition, each subject will be regularly assessed by the medical staff throughout the clinical trial and whenever the investigator deems necessary. As a minimum, subjects will be questioned for AEs (and concomitant therapies) at the time points indicated in the <u>Flow Chart</u>. Assessment will be made using non-specific questions such as 'How do you feel?'. Specific questions will be asked wherever necessary in order to more precisely describe an AE.

A carefully written record of all AEs shall be kept by the investigator in charge of the trial. Records of AEs shall include data on the time of onset, end time, intensity of the event, and any treatment or action required for the event and its outcome.

The following must be collected and documented on the appropriate CRF(s) by the investigator:

- From signing the informed consent onwards until an individual subject's end of trial (the End of Study (EoS) visit):
  - o All AEs (serious and non-serious) and all AESIs
  - The only exception to this rule are AEs (serious and non-serious) and AESIs
    in Phase I trials in healthy volunteers, when subjects discontinue from the trial
    due to screening failures prior to administration of any trial medication. In

c36231686-05

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

these cases, the subjects' data must be collected at trial site but will not be entered in the CRF and will not be reported in the CTR.

- After the individual subject's end of trial:
  - o The investigator does not need to actively monitor the subject for new AEs but should only report any occurrence of cancer and trial treatment related SAEs and trial treatment related AESIs of which the investigator may become aware of by any means of communication, e.g. phone call. Those AEs should be reported on the BI SAE form (see Section 5.2.6.2.2), but not on the CRF.

#### 5.2.6.2.2 AE reporting to the sponsor and timelines

The Investigator must report SAEs, AESIs, and non-serious AEs which are relevant for the reported SAE or AESI, on the BI SAE form to the sponsor's unique entry point immediately (without undue delay) The country specific reporting process (contact details) will be provided in the ISF. The same timeline applies if follow-up information becomes available. On specific occasions, the Investigator could inform the sponsor upfront via telephone. This does not replace the requirement to complete and send the BI SAE form.

With receipt of any further information to these events, a follow-up SAE form has to be provided. For follow-up information, the same rules and timeline apply as for initial information. All (S)AEs, including those persisting after the individual subject's end of trial, must be followed up until they have resolved, have been sufficiently characterized (e.g. as 'chronic' or 'stable'), or no further information can be obtained.

#### 5.2.6.2.3 Pregnancy

In rare cases, pregnancy might occur in a clinical trial. Once a subject has been enrolled in the clinical trial and has taken trial medication, the investigator must report any drug exposure during pregnancy in a trial participant immediately (within 24 hours) by means of Part A of the Pregnancy Monitoring Form to the sponsor's unique entry point.

The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported to the sponsor's unique entry point on the Pregnancy Monitoring Form for Clinical Studies (Part B). The ISF will contain the Pregnancy Monitoring Form for Clinical Studies (Part A and Part B).

As pregnancy itself is not to be reported as an AE, in the absence of an accompanying SAE and/or AESI, only the Pregnancy Monitoring Form for Clinical Studies and not the SAE form is to be completed. If there is an SAE and/or AESI associated with the pregnancy, an SAE form must be completed in addition.

#### 5.2.6.2.4 AE reporting from suicidality assessment

All positive reports from C-SSRS suicidality assessment (see section <u>5.2.5.1</u>), i.e. reports of suicidal ideation type 4 or 5 and all reports of suicidal behaviour must be reported as separate SAEs by the investigator.


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Negative reports (i.e. suicidal ideation type 1, 2 or 3) can be reported as AEs, at the discretion of the investigator. All negative reports should be reviewed by the Investigator for clinical relevance and determination if an AE report is warranted.

### 5.3 DRUG CONCENTRATION MEASUREMENTS AND PHARMACOKINETICS

#### 5.3.1 Assessment of pharmacokinetics

For the assessment of pharmacokinetics, blood samples will be collected at the time points indicated in the <u>Flow Chart</u>. The actual sampling times will be recorded and used for determination of pharmacokinetic parameters.

#### 5.3.2 Methods of sample collection

#### 5.3.2.1 Blood sampling for pharmacokinetic analysis

For quantification of BI 1358894 concentrations in plasma, 2.7 mL of blood will be drawn from an antecubital or forearm vein into an K<sub>2</sub>-EDTA (dipotassium ethylenediaminetetraacetic acid)-anticoagulant blood drawing tube at the times indicated in the Flow Chart. Blood will be withdrawn by means of either an indwelling venous catheter or by venipuncture with a metal needle.

The EDTA-anticoagulated blood samples will be centrifuged for approximately 10 min at approximately 2000 g to 4000 g and at 4 to 8 °C. Two plasma aliquots will be obtained and stored in polypropylene tubes. The first aliquot should contain at least 0.5 mL of plasma. The process from blood collection until transfer of plasma aliquots into the freezer should be completed within 120 minutes, with interim storage of blood samples and aliquots at room temperature. The time each aliquot was placed in the freezer will be documented. Until transfer on dry ice to the analytical laboratory, the aliquots will be stored upright at approximately -20°C or below at the trial site. The second aliquot will be transferred to the analytical laboratory after the bioanalyst has acknowledged safe arrival of the first aliquot. At the analytical laboratory, the plasma samples will be stored at approximately -20°C or below until analysis.

At a minimum, the sample tube labels should list BI trial number, subject number, visit, and planned sampling time.

After analysis, the plasma samples may be used for further methodological investigations (e.g. for stability testing or assessment of metabolites) or to address Health Authority questions regarding the results/methodology. However, only data related to the analyte and/or its metabolite(s) including anti-drug antibodies (if applicable) will be generated by these additional investigations. The trial samples will be discarded after completion of the additional investigations but not later than 5 years after the CTR is archived.



#### 5.3.4 Pharmacokinetic - pharmacodynamic relationship

No analysis of the relationship between pharmacokinetic and pharmacodynamic parameters is planned for this trial.

#### 5.4 ASSESSMENT OF BIOMARKERS

Not applicable

#### 5.5 BIOBANKING

Not applicable.

#### 5.6 OTHER ASSESSMENTS

#### 5.6.1 Pharmacogenomic evaluation

Pharmacogenomic investigations explore the role of genetic variation in determining an individual's response to drugs. For this purpose, a sample of at most 10 mL of blood will be obtained at the screening examination from each subject whose genotype has not been previously determined. Separate informed consent for genotyping will be obtained from each volunteer prior to sampling.

Deoxyribonucleic acid (DNA) will be extracted from the blood sample in order to sequence genes coding for proteins that are involved in the absorption, distribution, metabolism, and excretion (ADME) of drugs. The gene sequences to be determined include known and likely functional variations of key ADME genes and incorporate more than 90% of ADME-related genetic markers identified by the PharmaADME group (weblink ). It is not intended to include the pharmacogenomic data in the CTR. However, the data may be part of the CTR, if necessary.

#### 5.7 APPROPRIATENESS OF MEASUREMENTS

All measurements performed during this trial are standard measurements and will be performed in order to monitor subjects' safety and to determine pharmacokinetic parameters in an appropriate way.

The scheduled measurements will allow monitoring of changes in vital signs and standard laboratory values that might occur as a result of administration of trial medication. The safety

Boehringer Ingelheim BI Trial No.: 1402-0020

**Trial Protocol** 

c36231686-05

eim 20 Apr 2022


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

assessments are standard, are accepted for evaluation of safety and tolerability of an orally administered drug, and are widely used in clinical trials. The pharmacokinetic parameters and measurements outlined in Section 5.3 are generally used assessments of drug exposure. Prospective suicidality assessment is performed in this trial using the recommended C-SSRS questionnaire [R08-1147, R12-4395]

**c36231686-05** Trial Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6. INVESTIGATIONAL PLAN

#### 6.1 VISIT SCHEDULE

Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening and the end of trial examination are provided in the Flow Chart.

Study measurements and assessments scheduled to occur 'before' trial medication administration on Day 1 are to be performed and completed within a 3 h-period prior to the trial drug administration.

Up to 48 h after drug administration (planned time), the acceptable deviation from the scheduled time for adverse event/concomitant medication questioning, suicidality assessment, vital signs, ECG, and laboratory tests will be  $\pm$  30 min, if not stated otherwise in the Flow Chart,

For PK sampling, no time window is defined for this period (i.e. up to 48 h after drug administration).

Starting from planned time of 48 hours after drug administration (and beyond) a time window of +/- 120 minutes will be allowed for all procedures

Starting from a planned time of 168 hours after drug administration (and beyond) a time window of  $\pm$ 0 hours will be allowed for all procedures

If scheduled in the Flow Chart at the same time as a meal, blood sampling, vital signs, and 12-lead ECG recordings have to be done first. Furthermore, if several measurements including venipuncture are scheduled for the same time, venipuncture should be the last of the measurements due to its inconvenience to the subject and possible influence on physiological parameters.

For planned blood sampling times, refer to the Flow Chart. While these nominal times should be adhered to as closely as possible, the actual sampling times will be recorded and used for the determination of pharmacokinetic parameters.

If a subject misses an appointment, it will be rescheduled if possible. The relevance of measurements outside the permitted time windows will be assessed no later than at the Report Planning Meeting.

#### 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

#### 6.2.1 Screening

After having been informed about the trial, all subjects will provide written informed consent in accordance with GCP and local legislation prior to enrolment in the trial.

For information regarding laboratory tests (including drug and virus screening), ECG, vital signs, suicidality assessment, and physical examination, refer to Sections 5.2.1 to 5.2.5.

Genotyping will be performed in those volunteers whose genotypes have not been previously determined (for details, see Section 5.6).

At Screening, adequate contraceptive measures are described and the background why strict adherence to the measures is required.

It must be reiterated, at all visits following a screening, that WOCBP are using the appropriate method of safe contraception pursuant to section 4.2.2.3.

#### 6.2.2 Treatment period

Each subject is expected to participate in 4 treatment periods (each consisting of Days -1, 1-7, 11 and 14 in each period). At least 17 days will separate drug administrations in the first, second, third and fourth treatment period.

In the evening of Day -1 of each treatment period, trial participants will be admitted to the trial site and kept under close medical surveillance for at least 24 hours following drug administration. The subjects will then be allowed to leave the trial site after formal assessment and confirmation of their fitness. On all other trial days, subjects will be treated in an ambulatory fashion.

For details on time points and procedures for collection of plasma samples for PK analysis, refer to Flow Chart and Section 5.3.2.

The safety measurements performed during the treatment period are specified in Section <u>5.2</u> of this protocol and in the Flow Chart. AEs and concomitant therapy will be assessed continuously from obtaining subject's written informed consent until the end of trial examination. For details on times of all other trial procedures, refer to the Flow Chart.

#### 6.2.3 Follow-up period and trial completion

For AE assessment, laboratory tests, suicidality assessment, recording of ECG and vital signs, and physical examination during the follow-up period, see Section 5.2.

Subjects who discontinue treatment before the end of the planned treatment period should undergo the EoS Visit.

If needed in the opinion of the investigator, additional visits may be scheduled after the EoS Visit for continued safety monitoring.

All abnormal values (including laboratory parameters) that are assessed as clinically relevant by the investigator will be monitored using the appropriate tests until a return to a medically acceptable level is achieved. (S)AEs persisting after a subject's EoS Visit must be followed until they have resolved, have been sufficiently characterised, or no further information can be obtained.

20 Apr 2022

C36231686-05 Trial Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

#### 7.1 NULL AND ALTERNATIVE HYPOTHESES

The relative bioavailability of the interested treatment comparisons:

- i) T<sub>fasted</sub> versus R<sub>fasted</sub>
- ii) T<sub>fed</sub> versus R<sub>fed</sub>
- iii) T<sub>fed</sub> versus T<sub>fasted</sub>
- iv) R<sub>fed</sub> versus R<sub>fasted</sub>

will be estimated by the ratios of the geometric means (treatment A/treatment B, with A, B representing first, respectively second treatment of each pairwise comparisons stated above), and their corresponding 2-sided 90% confidence intervals (CIs) will be provided. This method corresponds to the two one-sided t-test procedure, each at the 5% significance level. Since the main focus is on estimation and not testing, a formal hypothesis test and associated acceptance range is not specified.

Due to the exploratory nature of the assessment, no significance level adjustment for investigating multiple comparisons will be applied.

#### 7.2 PLANNED ANALYSES

#### 7.2.1 General considerations

#### 7.2.1.1 Analysis sets

Statistical analyses will be based on the following analysis sets:

- Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug. The treated set will be used for safety analyses.
- Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability (as specified in the following subsection 'Pharmacokinetics'). Thus, a subject will be included in the PKS, even if he/she contributes only one PK parameter value for one period to the statistical assessment. Descriptive and model-based analyses of PK parameters will be based on the PKS.

Descriptions of additional analysis sets may be provided in the TSAP.

Adherence to the protocol will be assessed by the trial team. Important protocol deviation (iPD) categories will be suggested in the iPD specification file. IPDs will be identified no later than in the Report Planning Meeting, and the iPD categories will be updated as needed.

#### 7.2.1.2 Pharmacokinetics

The pharmacokinetic parameters listed in Section 2.1 and 2.2.2 for drug BI 1358894 will be calculated according to the relevant BI internal procedures.

Plasma concentration data and parameters of a subject will be included in the statistical pharmacokinetic (PK) analyses if they are not flagged for exclusion due to a protocol deviation relevant to the evaluation of PK (to be decided no later than in the Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the CTR.

Important protocol deviations may be

- Incorrect trial medication taken, i.e. the subject received at least one dose of trial medication the subject was not assigned to
- Incorrect dose of trial medication taken
- Incorrect intake of meal prior to drug administration in treatment periods under fed condition
- Use of restricted medications

Plasma concentrations and/or parameters of a subject will be considered as non-evaluable, if for example

- The subject experienced emesis that occurred at or before two times median t<sub>max</sub> of the respective treatment (Median t<sub>max</sub> is to be determined excluding the subjects experiencing emesis),
- A BI 1358894 predose concentration is >5% C<sub>max</sub> value for a subject for a specific treatment period, that specific treatment period will be excluded
- Missing samples/concentration data at important phases of PK disposition curve

Plasma concentration data and parameters of a subject which are flagged for exclusion will be reported with its individual values but will not be included in the statistical analyses. Descriptive and inferential statistics of PK parameters will be based on the PKS.

Only concentration values within the validated concentration range and actual sampling times will be used for the calculation of pharmacokinetic parameters. Concentrations used in the pharmacokinetic calculations will be in the same format provided in the bioanalytical report, (that is, to the same number of decimal places provided in the bioanalytical report).

#### 7.2.2 Primary endpoint analyses

#### Primary analyses

The statistical model used for the analysis of the primary endpoints will be an analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoints will be log-transformed (natural logarithm) prior to fitting the ANOVA model. This model will include effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment.

The effect 'subjects within sequences' will be considered as random, whereas the other effects will be considered as fixed. The model is described by the following equation:

$$y_{ijkm} = \mu + \zeta_i + s_{im} + \pi_j + \tau_k + e_{ijkm}$$
, where

 $y_{ijkm}$  = logarithm of response measured on subject m in sequence i receiving treatment k in period j,

 $\mu$  = the overall mean,

 $\zeta_i$  = the i<sup>th</sup> sequence effect, i = 1, 2, 3, 4

 $s_{im}$  = the effect associated with the  $m^{th}$  subject in the  $i^{th}$  sequence, m = 1, 2, ..., 6

 $\pi_i$  = the j<sup>th</sup> period effect, j = 1, 2, 3, 4

 $\tau_k$  = the k<sup>th</sup> treatment effect, k = 1, 2, 3, 4

 $e_{ijkm}$  = the random error associated with the  $m^{th}$  subject in sequence i who received treatment k in period j.

where  $s_{im} \sim N(0, \sigma_B^2)$  i.i.d.,  $e_{ijkm} \sim N(0, \sigma_W^2)$  i.i.d. and  $s_{im}$ ,  $e_{ijkm}$  are independent random variables.

Point estimates for the ratios of the geometric means (treatment A / treatment B) for the comparisons as stated in Section  $\underline{7.1}$  and the primary endpoints (see Section  $\underline{2.1}$ ) with their two-sided 90% confidence intervals (CIs) will be provided.

For each endpoint, the difference between the expected means for log(A)-log(B) will be estimated by the difference in the corresponding adjusted means (Least Squares Means). Additionally, their two-sided 90% confidence intervals will be calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint.

#### 7.2.3 Secondary endpoint analyses

The secondary endpoint (refer to Section 2.1.3) will be calculated according to the relevant BI internal procedures and will be assessed statistically using the same methods as described for the primary endpoints.


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 7.2.5 Safety analyses

Safety will be analysed based on the assessments described in Section <u>2.2.2.2</u>. All treated subjects (TS, refer to Section <u>7.2</u>) will be included in the safety analysis. Safety analyses will be descriptive in nature and based on BI standards. No hypothesis testing is planned.

For all analyses, the treatment actually administered (= treatment at onset) to the subject will be used (any deviations from the randomised treatment will be discussed in the minutes of the Report Planning Meeting).

Treatments will be compared in a descriptive way. Tabulations of frequencies/proportions will be used to evaluate categorical (qualitative) data, and tabulations of descriptive statistics will be used to analyse continuous (quantitative) data.

Measurements (such as ECG, vital signs, or laboratory parameters) or AEs will be assigned to treatments (see Section 4.1) based on the actual treatment at the time of the measurement or on the recorded time of AE onset (concept of treatment emergent AEs). Therefore, measurements performed or AEs recorded prior to first intake of trial medication will be assigned to the screening period, those between first trial medication intake and end of REP (see Section 1.2.2) will be assigned to the respective treatment period. Events occurring after the REP but prior to next intake or end of trial termination date will be assigned to 'follow-up'. In case of two or more treatments, the follow-up will be summarized according to the previous treatment. These assignments including the corresponding time intervals will be defined in detail in the TSAP. Note that AEs occurring after the last per protocol contact but entered before final database lock will be reported to Pharmacovigilance only and will not be captured in the trial database.

Additionally, further treatment intervals (analysing treatments) may be defined in the TSAP in order to provide summary statistics for time intervals, such as combined treatments, ontreatment totals, or periods without treatment effects (such as screening and follow-up intervals).

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Frequency, severity, and causal relationship of AEs will be tabulated by treatment, system organ class, and preferred term. SAEs, AESIs (see Section <u>5.2.6.1</u>), and other significant AEs (according to ICH E3) will be listed separately.

Relevant ECG findings will be reported as AEs.

Reports of C-SSRS will be reported as AEs as described in Section <u>5.2.6.2.4</u> and will be summarized as such. Results of the C-SSRS will be provided as listing.

Previous and concomitant therapies will be presented per treatment sequence group.

c36231686-05 Trial Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Laboratory data will be compared to their reference ranges. Values outside the reference range as well as possibly clinically significant values will be highlighted in the listings. Additionally, differences from baseline will be evaluated.

Vital signs or other safety-relevant data will be assessed with regard to possible on-treatment changes from baseline.

#### 7.2.6 Interim analyses

No interim analysis is planned.

#### 7.3 HANDLING OF MISSING DATA

#### **7.3.1** Safety

It is not planned to impute missing values for safety parameters.

#### 7.3.2 Pharmacokinetics

Handling of missing PK data will be performed according to the relevant BI internal procedures.

PK parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed.

#### 7.4 RANDOMISATION

Subjects will be randomised to one of the 4 treatment sequences in a 1:1:1:1 ratio. The block size will be documented in the CTR.

The sponsor will arrange for the randomisation as well as packaging and labelling of trial medication. The randomisation scheme will be generated using a validated system that uses a pseudo-random number generator and a supplied seed number so that the resulting allocation is both reproducible and non-predictable.

The randomisation scheme will contain additional blocks to allow for subject replacement (refer to Section 3.3.5).

#### 7.5 DETERMINATION OF SAMPLE SIZE

It is planned to enter a total of 24 subjects in the trial including up to 4 drop-outs. The sample size is considered sufficient to achieve the aims of this exploratory trial. With this sample size, the following precision in estimating the ratio of geometric means (treatment A/ treatment B; with A, B representing respective treatments of the pairwise treatment comparisons of interest, see Section 7.1) can be expected with 95% probability. Precision is defined as the ratio of upper CI limit (CL) to the relative BA estimate. Note that the precision is independent of the actual ratio of geometric means.

The observed intra-individual coefficient of variation (gCV) for BI 1358894 TFII in previous trial (1402-0010 [c28907328]) was roughly 25% for  $C_{max}$  and 13% for AUC.

For various assumptions around the gCV of 15-25%, Table 7.5: 1 provides an overview of the achievable precision for estimating the ratio of geometric means (treatment A/treatment B) for the formulation differences, i.e. comparisons i) and ii) (see Section 7.1). Table 7.5: 2 provides an overview of the achievable precision for estimating the food effect of each formulation, i.e. comparisons iii) and iv) (see Section 7.1),

. For illustrative purposes, the expected 90% confidence intervals are displayed for different values of the ratios A/B of geometric means. Note, as the same intra-individual gCVs and sample sizes N are assumed for the assessment of formulation differences and food effect, the precisions in Table 7.5.1 and 7.5.2 are the same, only different ratios are expected and are displayed with the respective 90% CI in the tables below.

Table 7.5: 1 Precision that can be expected with 95% probability and illustrative two-sided 90% confidence intervals around the ratios of geometric means (A/B) for different gCVs in a 4x4 crossover trial (N=20, 24) assessing formulation differences

| N | gCV<br>[%] | Precision<br>upper CL** / | 90% C | I [%] of respectiv | e ratio* |
|---|---|---|---|---|---|
| | [70] | relative BA<br>estimate | 90 | 100 | 110 |
| | 15 | 1.10 | (82.15; 98.60) | (91.23; 109.56) | (100.41; 120.51) |
| 20 | 20 | 1.13 | (79.73; 101.59) | (88.59; 112.88) | (97.45; 124.17) |
| | 25 | 1.16 | (77.42; 104.63) | (86.02; 110.44) | (94.62; 127.88) |
| | 15 | 1.09 | (82.92; 97.69) | (92.13; 108.54) | (101.34; 119.40) |
| 24 | 20 | 1.12 | (80.72; 100.35) | (89.69; 111.50) | (98.66; 122.65) |
| | 25 | 1.15 | (78.61; 103.04) | (87.34; 114.49) | (96.08; 125.94) |

<sup>\*</sup>Ratio of geometric means (A/B) for a PK endpoint is defined by exp(µA)/exp(µB)

<sup>\*\*</sup>Confidence interval limit

c36231686-05

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.5: 2 Precision that can be expected with 95% probability and illustrative two-sided 90% confidence intervals around the ratios of geometric means (A/B) for different gCVs in a 4x4 crossover trial (N=20, 24) assessing food effect

| gCV | Precision | 90% C | I [%] of respectiv | e ratio* |
|---|---|---|---|---|
| [70] | relative BA<br>estimate | 100 | 115 | 180 |
| 15 | 1.10 | (91.23; 109.56) | (104.97; 125.99) | (164.30; 197.20) |
| 20 | 1.13 | (88.59; 112.88) | (101.88; 129.81) | (159.46; 203.18) |
| 25 | 1.16 | (86.02; 110.44) | (98.92; 133.70) | (154.83; 209.26) |
| 15 | 1.09 | (92.13; 108.54) | (105.95; 124.83) | (165.83; 195.38) |
| 20 | 1.12 | (89.69; 111.50) | (103.14; 128.22) | (161.44; 200.70) |
| 25 | 1.15 | (87.34; 114.49) | (100.44; 131.67) | (157.22; 206.08) |
| | [%] 15 20 25 15 20 | [%] upper CL** / relative BA estimate 15 | wpper CL**/ relative BA estimate | [%] upper CL**/relative BA estimate 100 115 15 1.10 (91.23; 109.56) (104.97; 125.99) 20 1.13 (88.59; 112.88) (101.88; 129.81) 25 1.16 (86.02; 110.44) (98.92; 133.70) 15 1.09 (92.13; 108.54) (105.95; 124.83) 20 1.12 (89.69; 111.50) (103.14; 128.22) |

<sup>\*</sup>Ratio of geometric means (A/B) for a PK endpoint is defined by  $\exp(\mu_A)/\exp(\mu_B)$ .

The expected 90% confidence interval limits in the tables above were derived by

CI limit<sub>upper.lower</sub> = 
$$\exp(\ln(\theta) \pm \omega)$$
,

with  $\theta$  being the ratio (A/B) on original scale and  $\omega$  the distance from the estimate  $\theta$  to either confidence interval limit on the log-scale, which was obtained from the achievable precision on the original scale.

The calculation was performed as described by Julious [R11-5230] using R Version 4.0.2.

<sup>\*\*</sup>Confidence interval limit

**Trial Protocol** 

c36231686-05

20 Apr 2022


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8. INFORMED CONSENT, TRIAL RECORDS, DATA PROTECTION, PUBLICATION POLICY, AND ADMINISTRATIVE STRUCTURE

The trial will be carried out in compliance with the protocol, the ethical principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonized Guideline for Good Clinical Practice (GCP), relevant BI Standard Operating Procedures (SOPs), the EU directive 2001/20/EC, and other relevant regulations. Investigators and site staff must adhere to these principles. Deviation from the protocol, the principles of ICH GCP or applicable regulations will be treated as 'protocol deviation'.

Standard medical care (prophylactic, diagnostic, and therapeutic procedures) remains the responsibility of the subject's treating physician.

The investigator will inform the sponsor immediately of any urgent safety measures taken to protect the trial subjects against any immediate hazard, as well as of any serious breaches of the protocol or of ICH GCP.

The Boehringer Ingelheim transparency and publication policy can be found on the following web page: trials.boehringer-ingelheim.com. As a general rule, no trial results should be published prior to finalisation of the CTR.

The terms and conditions of the insurance coverage are made available to the investigator and the subjects and are stored in the ISF.

#### 8.1 TRIAL APPROVAL, SUBJECT INFORMATION, INFORMED CONSENT

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB / Independent Ethics Committee (IEC and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments. Prior to a subject's participation in the trial, written informed consent must be obtained from each subject (or the subject's legally accepted representative) according to ICH-GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional subject-information form retained by the investigator as part of the trial records. A signed copy of the informed consent and any additional subject information must be given to each subject or the subject's legally accepted representative.

The subject must be given sufficient time to consider participation in the trial. The investigator or delegate obtains written consent of the subject's own free will with the informed consent form after confirming that the subject understands the contents. The investigator or delegate must sign (or place a seal on) and date the informed consent form. If a trial collaborator has given a supplementary explanation, the trial collaborator also signs (or places a seal on) and dates the informed consent.

Re-consenting may become necessary when new relevant information becomes available and should be conducted according to the sponsor's instructions.

The consent and re-consenting process should be properly documented in the source documentation.

For subjects enrolled during the COVID-19 pandemic: In addition to the study-specific informed consent, separate written consent will be obtained for testing for SARS-CoV-2 infection.

#### 8.2 DATA QUALITY ASSURANCE

A risk-based approach is used for trial quality management. It is initiated by the assessment of critical data and processes for trial subject protection and reliability of the results as well as identification and assessment of associated risks. An Integrated Quality and Risk Management Plan or alternative plan, in line with the guidance provided by ICH Q9 and ICH-GCP E6, for fully outsourced trials, documents the rationale and strategies for risk management during trial conduct including monitoring approaches, vendor management and other processes focusing on areas of greatest risk.

Continuous risk review and assessment may lead to adjustments in trial conduct, trial design or monitoring approaches.

A quality assurance audit/inspection of this trial may be conducted by the sponsor, sponsor's designees, or by IRB / IEC or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial.

#### 8.3 RECORDS

CRFs for individual subjects will be provided by the sponsor. For drug accountability, refer to Section 4.1.8.

#### 8.3.1 Source documents

In accordance with regulatory requirements, the investigator should prepare and maintain adequate and accurate source documents and trial records for each trial subject that include all observations and other data pertinent to the investigation. Source data as well as reported data should follow the 'ALCOA principles' and be <u>attributable</u>, <u>legible</u>, <u>contemporaneous</u>, <u>original</u>, and <u>accurate</u>. Changes to the data should be traceable (audit trail).

Data reported on the CRF must be consistent with the source data or the discrepancies must be explained.

The current medical history of the subject may not be sufficient to confirm eligibility for the trial and the investigator may need to request previous medical histories and evidence of any diagnostic tests. In this case, the investigator must make at least one documented attempt to retrieve previous medical records. If this fails, a verbal history from the subject, documented in their medical records, would be acceptable.

Before providing any copy of subjects' source documents to the sponsor, the investigator must ensure that all subject identifiers (e.g., subject's name, initials, address, phone number, and social security number) have properly been removed or redacted to ensure subject confidentiality.

If the subject is not compliant with the protocol, any corrective action (e.g. re-training) must be documented in the subject file.

For the CRF, data must be derived from source documents, for example:

- Subject identification: gender, year of birth (in accordance with local laws and regulations)
- Subject participation in the trial (substance, trial number, subject number, date subject was informed)
- Dates of subject's visits, including dispensing of trial medication
- Medical history (including trial indication and concomitant diseases, if applicable)
- Medication history
- AEs and outcome events (onset date [mandatory], and end date [if available])
- SAEs (onset date [mandatory], and end date [if available])
- Concomitant therapy (start date, changes)
- Originals or copies of laboratory results and other imaging or testing results, with proper documented medical evaluation (in validated electronic format, if available)
- ECG results (original or copies of printouts)
- Completion of subject's participation in the trial (end date; in case of premature discontinuation, document the reason for it, if known)
- Prior to allocation of a subject to a treatment into a clinical trial, there must be
  documented evidence in the source data (e.g. medical records) that the trial participant
  meets all inclusion criteria and does not meet any exclusion criteria. The absence of
  records (either medical records, verbal documented feedback of the subject or testing
  conducted specific for a protocol) to support inclusion/exclusion criteria does not
  make the subject eligible for the clinical trial.
- C-SSRS questionnaires

Data directly entered into ClinBase<sup>TM</sup> (that is, without prior written or electronic record) are considered to be source data. The place where data are entered first will be defined in a trial specific Source Data Agreement. The data in ClinBase<sup>TM</sup> are available for inspection at any time.


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8.3.2 Direct access to source data and documents

The investigator/institution will allow site trial-related monitoring, audits, IRB / IEC review and regulatory inspections. Direct access must be provided to the CRF and all source documents/data, including progress notes, copies of laboratory and medical test results, which must be available at all times for review by the Clinical Research Associate, auditor and regulatory inspector (e.g. FDA). They may review all CRFs and informed consents. The accuracy of the data will be verified by direct comparison with the source documents described in Section 8.3.1. The sponsor will also monitor compliance with the protocol and GCP.

#### 8.3.3 Storage period of records

#### Trial site:

The trial site must retain the source and essential documents (including ISF) according to the local requirements valid at the time of the end of the trial.

#### Sponsor:

The sponsor must retain the essential documents according to the sponsor's SOPs.

#### 8.4 EXPEDITED REPORTING OF ADVERSE EVENTS

BI is responsible to fulfil their legal and regulatory reporting obligation in accordance with regulatory requirements.

#### 8.5 STATEMENT OF CONFIDENTIALITY AND SUBJECT PRIVACY

Data protection and data security measures are implemented for the collection, storage and processing of subject data in accordance with the principles 7 and 12 of the WHO GCP handbook.

Individual subject data obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited with the following exceptions:

Personalised treatment data may be given to the subject's personal physician or to other appropriate medical personnel responsible for the subject's welfare. Data generated at the site as a result of the trial need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB / IEC and the regulatory authorities.

### 8.5.1 Collection, storage and future use of biological samples and corresponding data

Measures are in place to comply with the applicable rules for the collection, storage and future use of biological samples and clinical data, in particular

- Sample and data usage have to be in accordance with the informed consent
- The BI-internal facilities storing biological samples from clinical trial participants as well as the external storage facility are qualified for the storage of biological samples collected in clinical trials.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- An appropriate sample and data management system, incl. audit trail for clinical data and samples to identify and destroy such samples according to ICF is in place
- A fit for the purpose documentation (e.g. biomarker proposal, analysis plan and report) ensures compliant usage
- A fit for purpose approach will be used for assay/equipment validation depending on the intended use of the biomarker data
- Samples and/or data may be transferred to third parties and other countries as specified in the ICF

#### 8.6 TRIAL MILESTONES

The <u>start of the trial</u> is defined as the date when the first subject in the whole trial signs informed consent.

The <u>end of the trial</u> is defined as the date of the last visit of the last subject in the whole trial ('Last Subject Completed').

<u>Early termination of the trial</u> is defined as the premature termination of the trial due to any reason before the end of the trial as specified in this protocol.

<u>Temporary halt of the trial</u> is defined as any unplanned interruption of the trial by the sponsor with the intention to resume it.

<u>Suspension of the trial</u> is defined as an interruption of the trial based on a Health Authority request.

The IEC / competent authority in each participating EU member state will be notified about the trial milestones according to the laws of each member state.

A final report of the clinical trial data will be written only after all subjects have completed the trial in all countries (EU or non-EU), so that all data can be incorporated and considered in the report.

#### 8.7 ADMINISTRATIVE STRUCTURE OF THE TRIAL

The trial is sponsored by Boehringer Ingelheim (BI).

The trial will be conducted at the description of BI Pharma GmbH & Co. KG, Biberach, Germany, under the supervision of the Principal Investigator. Relevant documentation on the participating (Principal) Investigators (e.g. their curricula vitae) will be filed in the ISF. The investigators will have access to the BI web portal Clinergize to access documents provided by the sponsor.

BI has appointed a Clinical Trial Leader (CT Leader), responsible for coordinating all required trial activities, in order to

- Manage the trial in accordance with applicable regulations and internal SOPs
- Direct the clinical trial team in the preparation, conduct, and reporting of the trial

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

 Ensure appropriate training and information of local Clinical Trial Managers (CT Managers), Clinical Research Associates (CRAs), and investigators of participating trial sites

| The trial medication will be provided by the |
|---|
| · |
| Safety laboratory tests will be performed by the local laboratory of the trial site ( |
| ). |
| Analyses of BI 1358894 concentrations in plasma will be performed at |
| · |

On-site monitoring will be performed by BI or a contract research organisation appointed by BI.

Data management and statistical evaluation will be done by BI or a contract research organisation according to BI SOPs.

Tasks and functions assigned in order to organise, manage, and evaluate the trial are defined according to BI SOPs. A list of responsible persons and relevant local information can be found in the ISF.


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. REFERENCES

#### 9.1 PUBLISHED REFERENCES

| P06-11895 | Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry 2006; 163(11); 1905-1917. |
|---|---|
| R03-2269 | Guidance for industry: food-effect bioavailability and fed bioequivalence studies. In: U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER) 2002:1-9. |
| R06-2872 | Trivedi MH, Rush AJ, Wisniewski SR, Warden D, McKinney W, Downing M, Berman SR, Farabaugh A, Luther JF, Nierenberg AA, Callan JA, Sackeim HA. Factors associated with health-related quality of life among outpatients with major depressive disorder: a STAR*D report. J Clin Psychiatry 2006; 67(2); 185-195. |
| R08-1147 | Posner K. State of the science: measurement of suicidal adverse events and the Columbia Suicide Severity Rating Scale. 47th NCDEU Ann Mtg, Boca Raton, 11 - 14 Jun 2007. 2007:15 |
| R08-4516 | Kessler RC, Chiu WT, Demler O, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV diorders in the national comorbidity survey replication. Arch Gen Psychiatry 2005; 62; 617-627. |
| R11-5230 | Julious SA. Sample sizes for clinical trials. Boca Raton: Taylor & Francis Group; 2010. |
| R12-4395 | Guidance for industry: suicidal ideation and behaviour: prospective assessment of occurrence in clinical trials (draft guidance, August 2012). web page: fda.gov/downloads/Drugs/GuidanceRegulatoryInformation/Guidances/UCM22 5130.pdf (access date: 5 October 2012); 2012. |
| R15-3888 | Riccio A, Li Y, Moon J, Kim KS, Smith KS, Rudolph U, Gapon S, Yao GL, Tsvetkov E, Rodig SJ, Veer A van't, Meloni EG, Carlezon WA, Bolshakov VY, Clapham DE. Essential role for TRPC5 in amygdala function and fear-related behavior. Cell 2009; 137(4); 761-772. |
| R15-4424 | American Psychiatric Association. Diagnostic and statistical manual of mental disorders (DSM-5). 5th ed.Arlington: American Psychiatric Association; 2013. |
| R16-5350 | Fowler MA, Sidiropoulou K, Ozkan ED, Phillips CW, Cooper DC. Corticolimbic expression of TRPC4 and TRPC5 channels in the rodent brain. Plos One 2007; 2(6); e573 |


| Proprietary confidenti | ial information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| R16-5472 | Koenigsberg HW, Denny BT, Fan J, Liu X, Guerreri S, Mayson SJ, et al. The neural correlates of anomalous habituation to negative emotional pictures in borderline and avoidant personality disorder patients. Am J Psychiatry 2014; 171(1); 82-90. |
| R16-5473 | Mandell D, Siegle G, Shutt L, Feldmiller J, Thase ME. Neural substrates of trait ruminations in depression. J Abnorm Psychol 2014; 123(1); 35-48. |
| R16-5474 | IsHak WW, Elbau I, Ismail A, Delaloye S, Ha K, Bolotaulo NI, et al. Quality of life in borderline personality disorder. Harvard Rev Psychiatry 2013; 21(3); 138-150. |
| R16-5475 | McClintock SM, Husain MM, Wisniewski SR, Nierenberg AA, Stewart JW, Trivedi MH, et al. Residual symptoms in depressed outpatients who respond by 50 % but do not remit to antidepressant medication. J Clin Psychopharmacol 2011; 31(2); 180-186. |
| R16-5476 | Links PS, Heslegrave R, Reekum R van. Prospective follow-up study of borderline personality disorder: prognosis, prediction of outcome, and axis II comorbidity. Can J Psychiatry 1998; 43(3); 265-270. |
| R16-5477 | Skodol AE, Siever LJ, Livesley WJ, Gunderson JG, Pfohl B, Widiger TA. The borderline diagnosis II: biology, genetics, and clinical course. Biol Psychiatry 2002; 51(12); 951-963. |
| R16-5483 | Ellison WD, Rosenstein L, Chelminski I, Dalrymple K, Zimmerman M. The clinical significance of single features of borderline personality disorder: anger, affective instability, impulsivity, and chronic emptiness in psychiatric outpatients. J Personal Disord 2016; 30(2); 261-270. |
| R21-1276 | Lee DJ, Schnitzlein CW, Wolf JP, Vythilingam M, Rasmusson AM, Hoge CW. Psychotherapy versus pharmacotherapy for posttraumatic stress disorder: systemic review and meta-analyses to determine first-line treatments. Depress Anxiety 2016; 33; 792-806. |
| R94-1529 | Chow SC, Liu JP. Design and analysis of bioavailability and bioequivalence studies. New York: Marcel Dekker Inc., 1992. |

#### 9.2 UNPUBLISHED REFERENCES

c10354149 . Investigator's Brochure BI 1358894 in Major Depressive Disorder and Borderline Personality Disorder. Current Version.

**Boehringer Ingelheim** BI Trial No.: 1402-0020

**Trial Protocol** 

20 Apr 2022

c36231686-05  Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Trial Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10. APPENDICES

#### 10.1 COLUMBA-SUICIDE SEVERITY RATING SCALE

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Baseline/Screening Version

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A, Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

| For reprints of the C-SSRS contact | 1051 Riverside Drive, New |
|---|---|
| York, New York, 10032; inquiries and training requirements contact | |
| © 2008 | |

C-SSRS Baseline Screening - United States/English - Mapi.

| Ask questions 1 and 2. If both are negative, proceed to "Suicida | | | | | |
|---|---|---|---|---|---|
| question 2 is "yes", ask questions 3, 4 and 5. If the answer to qu<br>"Intensity of Ideation" section below. | | He/SI | ne: Time<br>he Felt<br>Suicidal | Past<br>Mon | |
| 1. Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anymore, or wish Have you wished you were dead or wished you couldgo to sleep and not wake | | Yes | No | Yes | No 🗆 |
| If yes, describe: | | | | | |
| 2. Non-Specific Active Suicidal Thoughts General non-specific thoughts of wanting to end one's life/commit suicide (e.g., ways to kill oneself/associated methods, intent, or plan during the assessment pe | | Yes | No | Yes | No |
| If yes, describe: | | | | | |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) witho Subject endorses thoughts of suicide and has thought of at least one method durplan with time, place or method details worked out (e.g., thought of method to k say, "I thought about taking an overdose but I never made a specific plan as to never go through with it." Have you been thinking about how you might do this? | ing the assessment period. This is different than a specific<br>till self but not a specific plan). Includes person who would | Yes | No | Yes | No |
| If yes, describe: | | | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, without Sp Active suicidal thoughts of killing oneself and subject reports having some inter but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? | | Yes | No | Yes | No |
| If yes, describe: | | | | | |
| <ol> <li>Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and Have you started to work out or worked out the details of how to kill yourself?</li> </ol> | | Yes | No | Yes | No |
| If yes, describe: | | | | | |
| INTENSITY OF IDEATION | | | | | |
| The following features should be rated with respect to the most severe the least severe and 5 being the most severe). Ask about time he/she wa | | | | | |
| <u>Lifetime</u> - Most Severe Ideation: Type # (1-5) | | | | | st |
| B I I A I I I I I I I I I I I I I I I I | Description of Ideation | Most | Severe | Mo<br>Seve | 0000 |
| Past 12 Months - Most Severe Ideation: Type # (1-5) | Description of Ideation Description of Ideation | Most | Severe | 0.0000000 | 0000 |
| Type # (1-5) | | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week | Description of Ideation | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration | Description of Ideation | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week | Description of Ideation | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability | (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hour/s lot of time Controllability Could/can you stop thinking about killing yourself or wanting to a (1) Easily able to control thoughts with little difficulty | (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to (1) Easily able to control thoughts with little difficulty (3) Can control thoughts with some difficulty Deterrents | (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours'a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to a (1) Easily able to control thoughts with little difficulty (3) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty | (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to a (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty (3) Can control thoughts with some difficulty Are there things - anyone or anything (e.g., jamily, religion, pain acting on thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you | (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours'a lot of time Controllability Contidean you stop thinking about killing yourself or wanting to a (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty (3) Can control thoughts with some difficulty Deterrents Are there things - anyone or anything (e.g., family, religion, pain acting on thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you Reasons for Ideation | (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts of death) - that stopped you from wanting to die or (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (0) Does not apply | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to a (1) Easily able to control thoughts with little difficulty (3) Can control thoughts with some difficulty (3) Can control thoughts with some difficulty Deterrents Are there things - anyone or anything (e.g., family, religion, pain acting on thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents definitely stopped you Reasons for Ideation What sort of reasons did you have for thinking about wanting to a stop the way you were feeling (in other words you couldn't go on the stop the way you were feeling (in other words you couldn't go on the control was to the stop to the way you were feeling (in other words you couldn't go on the control was to the way you were feeling (in other words you couldn't go on the control was the control was to the way you were feeling (in other words you couldn't go on the control was to the control was the | (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts of death) - that stopped you from wanting to die or (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (6) Does not apply die or killing yourself? Was it to end the pain or living with this pain or how you were feeling) or | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to a (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty (3) Can control thoughts with some difficulty Are there things - anyone or anything (e.g., jamily, religion, pain acting on thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you Reasons for Ideation What sort of reasons did you have for thinking about wanting to a stop the way you were feeling (in other words you couldn't go on was it to get attention, revenge or a reaction from others? Or both | (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts of death) - that stopped you from wanting to die or (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (0) Does not apply die or killing yourself? Was it to end the pain or living with this pain or how you were feeling) or | Most | Severe | 0.0000000 | 0000 |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to a (1) Easily able to control thoughts with little difficulty (3) Can control thoughts with some difficulty (3) Can control thoughts with some difficulty Deterrents Are there things - anyone or anything (e.g., family, religion, pain acting on thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents definitely stopped you Reasons for Ideation What sort of reasons did you have for thinking about wanting to a stop the way you were feeling (in other words you couldn't go on the stop the way you were feeling (in other words you couldn't go on the control was to the stop to the way you were feeling (in other words you couldn't go on the control was to the way you were feeling (in other words you couldn't go on the control was the control was to the way you were feeling (in other words you couldn't go on the control was to the control was the | (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts of death) - that stopped you from wanting to die or (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (6) Does not apply die or killing yourself? Was it to end the pain or living with this pain or how you were feeling) or | Most | Severe | 0.0000000 | 0000 |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| SUICIDAL BEHAVIOR (Check all that apply, so long as these are separate events; must ask about all types) | | | | Past n.a.<br>Years | |
|---|---|---|---|---|---|
| Actual Attempt: | | | | Yes | No |
| A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as nonself. Intent does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered at attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger wh mouth but gun is broken so no injury results, this is considered an attempt. Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstance a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping fr a high floor/story). Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be infer Have you made a suicide attempt? | Yes | No | | | |
| Have you done anything to harm yourself? | | | F100 (W) | | |
| Have you done anything dangerous where you could have died? What did you do? | | | 1#of<br>mpts | Total<br>Atter | |
| Did youas a way to end your life? | | Auto | ampes | Auci | upts |
| Did you want to die (even a little) when you ? | | | _ | | _ |
| Were you trying to end your life when you? | | | | | |
| Or did you think it was possible you could have died from? | | | | | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress | , feel better, | | | | |
| get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) | | | | 100 | |
| If yes, describe: | | Yes | No | Yes | No |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | | | | |
| Interrupted Attempt: | | Yes | No | Yes | No |
| When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actually | ıl attempt | | | | |
| would have occurred). Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather tha attempt. Shooting: Person has gun pointed toward self gun is taken away by someone else, or is somehow prevented from pulli Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken ledge. Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. Has there been a time when you started to do something to end your life but someone or something stopped. | ng trigger.<br>down from | Total # of | | Total | |
| before you actually did anything? If yes, describe: | | inten | rupted | intern | iptea |
| Aborted Attempt: | | Yes | No | Yes | No |
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-<br>destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by<br>something else. | | | | | |
| Has there been a time when you started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe: | | | | Total<br>abor | |
| Duanaustany Asta au Dahaviani | | | | | _ |
| Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: | | | | Yes | No |
| 11 ) 90, 4004100. | | | | | |
| Suicidal Behavior: | | Yes | No | Yes | No |
| Suicidal behavior was present during the assessment period? | | | | | |
| Answer for Actual Attempts Only | Most Recent<br>Attempt<br>Date: | Most Lethal<br>Attempt<br>Date: | | Initial/Fi<br>Attempt<br>Date: | |
| Actual Lethality/Medical Damage: | Enter Code | Enter | Code | Enter ( | Code |
| O. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death | | _ | _ | | _ |
| Potential Lethality: Only Answer if Actual Lethality=0 | Enter Code | Enter | Code | Enter ( | Code |
| Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | | | | | |
| 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | | | - | - |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <a href="The Columbia Suicide History">The Columbia Suicide History</a>
Form, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact
York, New York, 10032; inquiries and training requirements contact
© 2008

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| SUICIDAL IDEATION | | |
|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suicidal Behavior" section. If the answer to question 2 is "yes", ask questions 3, 4 and 5. If the answer to question 1 and/or 2 is "yes", complete "Intensity of Ideation" section below. | 107.000 | e Last<br>isit |
| <ol> <li>Wish to be Dead</li> <li>Subject endorses thoughts about a wish to be dead or not alive anymore, or wish to fall asleep and not wake up.</li> <li>Have you wished you were dead or wished you could go to sleep and not wake up?</li> </ol> | Yes | No |
| If yes, describe: | | |
| 2. Non-Specific Active Suicidal Thoughts General, non-specific thoughts of wanting to end one's life/commit suicide (e.g., "T've thought about killing myself") without thoughts of ways to kill oneself/associated methods, intent, or plan during the assessment period. Have you actually had any thoughts of killing yourself? | Yes | No |
| If yes, describe: | _ | |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act<br>Subject endorses thoughts of suicide and has thought of at least one method during the assessment period. This is different than a specific plan with time,<br>place or method details worked out (e.g., thought of method to kill self but not a specific plan). Includes person who would say, "I thought about taking an<br>overdose but I never made a specific plan as to when, where or how I would actually do it and I would never go through with it."<br>Have you been thinking about how you might do this? | Yes | No |
| If yes, describe: | | |
| 4. Active Suicidal Ideation with Some Intent to Act, without Specific Plan Active suicidal thoughts of killing eneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: | Yes | No |
| | _ | |
| 5. Active Suicidal Ideation with Specific Plan and Intent<br>Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out.<br>Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? | Yes | No |
| If yes, describe: | | |
| INTENSITY OF IDEATION | _ | |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). | Τ., | |
| Most Severe Ideation: | 0.000 | ost<br>vere |
| Type# (1-5) Description of Ideation | | |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day | _ | |
| Duration | | |
| When you have the thoughts, how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous | _ | - |
| Controllability Could can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty (0) Does not attempt to control thoughts | - | _ |
| Deterrents Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to die or acting on thoughts of committing suicide? | - | _ |
| (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you (6) Deterrents definitely did not stop you (7) Deterrents definitely did not stop you (8) Does not apply | | |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| SUICIDAL BEHAVIOR | THE NAME OF | Last |
|---|---|---|
| (Check all that apply, so long as these are separate events; must ask about all types) | Vi | sit |
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as method to kill oneself. Intent | Yes | No |
| does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered an actual suicide attempt. There does not | | |
| have to be any injury or harm, just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no injury results, | | |
| this is considered an attempt. | | |
| Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstances. For example, a highly | | |
| lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window of a high floor/story). Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be inferred. | | |
| Have you made a suicide attempt? | | |
| Have you done anything to harm yourself? | | |
| Have you done anything dangerous where you could have died? | | # of |
| What did you do? | Atte | mpts |
| Did you as a way to end your life? | | |
| Did you want to die (even a little) when you? | _ | _ |
| Were you trying to end your life when you? | | |
| Or did you think it was possible you could have died from? | | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get | | |
| sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent). If yes, describe: | | |
| a yes weather. | Yes | No |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | |
| Interrupted Attempt: | | 190019 |
| When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have | Yes | No |
| occurred). Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. | | |
| Shooting: Person has gus mointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, | | |
| even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around | | |
| neck but has not yet started to hang - is stopped from doing so. | Total | # of |
| Has there been a time when you started to do something to end your life but someone or something stopped you before you | interr | upted |
| actually did anything? If yes, describe: | | |
| 11 765 1604104 | _ | _ |
| Aborted Attempt: | Yes | No |
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. | | |
| Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. | | |
| Has there been a time when you started to do something to try to end your life but you stopped yourself before you | Total | I# of |
| actually did anything? | | rted |
| If yes, describe: | | |
| Preparatory Acts or Behavior: | | _ |
| Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a | Yes | No |
| specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). | | |
| Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, | " | |
| giving valuables away or writing a suicide note)? | | |
| If yes, describe: | | |
| | Var | No |
| Suicidal Behavior: Suicidal behavior was present during the assessment period? | Yes | No |
| Solitions duration was problem during the association periods. | | |
| Suicide: | Yes | No |
| Answer for Actual Attempts Only | Most Le | |
| | Attempt<br>Date: | |
| Actual Lethality/Medical Damage: | Enter | 0.1. |
| No physical damage or very minor physical damage (e.g., surface scratches). | Enter | Coae |
| <ol> <li>Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains).</li> </ol> | | |
| <ol><li>Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel).</li></ol> | | |
| <ol> <li>Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns<br/>less than 20% of body; extensive blood loss but can recover; major fractures).</li> </ol> | | |
| 4. Severe physical damage, medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; | _ | _ |
| extensive blood loss with unstable vital signs; major damage to a vital area). | | |
| 5. Death | _ | |
| Potential Lethality: Only Answer if Actual Lethality=0 | Enter | Code |
| Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality; put gun in meuth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away | | |
| before an over). | | |
| 0 = Behavior not likely to result in injury | | |
| 1 = Behavior likely to result in injury but not likely to cause death | _ | _ |
| 2 = Behavior likely to result in death despite available medical care | I | |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11. DESCRIPTION OF GLOBAL AMENDMENTS

#### 11.1 GLOBAL AMENDMENT 1

| Date of amendment | | 15 Dec 2021 |
|---|---|---|
| EudraCT number | | 2021-004880-28 |
| EU number | | |
| BI Trial number | | 1402-0020 |
| BI Investigational Medicinal | | BI 1358894 |
| Product(s) | | |
| Title of protocol | | Relative bioavailability of two different tablet |
| | | formulations of BI 1358894 administered in healthy |
| | | subjects in fasted and fed state (an open-label, |
| | | randomised, single-dose, four-period, four-sequence |
| | | crossover study) |
| | 18 × | |
| Substantial Global Amendmen | nt du | e to urgent safety reasons |
| Substantial Global Amendment | | |
| Non-substantial Global Amendment | | |
| Section to be changed | 1. | Section 3.3.4.1 Withdrawal from trial treatment |
| | 2. | Section 3.3.4.3 Discontinuation of trial by the |
| | | sponsor |
| Description of change | 1. | Include an additional criterion for withdrawal of trial |
| | | treatment for an individual subject in case of severe |
| | | adverse drug reactions |
| | 2. | Include an additional criterion for discontinuation of |
| | | the trial in case of severe adverse drug reactions |
| D 4: 1 6 1 | 1 | TT 1/1 /1 // |
| Rationale for change | 1. | Health authority request |
| | 2 | Health outhority request |
| | 2. | Health authority request |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11.2 GLOBAL AMENDMENT 2

| Date of amendment | 11 Jan 2022 |
|---|---|
| EudraCT number | 2021-004880-28 |
| EU number | 2021 00 1000 20 |
| BI Trial number | 1402-0020 |
| BI Investigational Medicinal | BI 1358894 |
| Product(s) | |
| Title of protocol | Relative bioavailability of two different tablet |
| IIII of process | formulations of BI 1358894 administered in healthy |
| | subjects in fasted and fed state (an open-label, |
| | randomised, single-dose, four-period, four-sequence |
| | crossover study) |
| Substantial Global Amendmen | t due to urgent safety reasons |
| Substantial Global Amendment | |
| Non-substantial Global Amend | lment 🖂 |
| Non-substantial Global Ameno | |
| Section to be changed | 1. Section 5.2.5.1 |
| | 2. Section 10.1 |
| Description of change | 1. Deletion of one paragraph that appears identically |
| | at the end of the section |
| | 2. Columbia-Suicide Severity Rating Scale (C- |
| | SSRS) - Baseline/Screening version. |
| | a) Suicidal Ideation Assessment. |
| | The timeframe for 'most severe ideation' was |
| | changed from 6 months to 12 months. |
| | b) Suicidal Behavior Assessment |
| | In accordance to the original C-SSRS scale, a second |
| | column was inserted that would allow the |
| | assessment of suicidal behaviour for a pre-specified |
| | number of years. |
| | However, since a specific timeframe for suicidal |
| | behaviour is not evaluated in this trial, i.e. is not |
| | applicable, the header of the second column |
| D. (I. C. I. | contains the expression "Past n.a. years". |
| Rationale for change | 1. Correction |
| | 2. a) Correction |
| | 2. b) For transparency reasons and to ensure better |
| | consistency with the original C-SSRS |
| | Baseline/Screening Version |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11.3 GLOBAL AMENDMENT 3

| Date of amendment | 24 Jan 2022 |
|---|---|
| EudraCT number | 2021-004880-28 |
| EU number | |
| BI Trial number | 1402-0020 |
| BI Investigational Medicinal | BI 1358894 |
| Product(s) | |
| Title of protocol | Relative bioavailability of two different tablet formulations of BI 1358894 administered in healthy subjects in fasted and fed state (an open-label, randomised, single-dose, four-period, four-sequence |
| | crossover study) |
| Substantial Global Amendment due to urgent safety reasons | |
| Substantial Global Amendment | |
| Non-substantial Global Amendment | |
| | To a series and a |
| Section to be changed | 5.2.3. Safety laboratory |
| Description of change | In line with the current Investigator's Brochure |
| | (section 7.6.1) sexual hormones (total testosterone, |
| | FSH, LH) shall be performed in males only. |
| Rationale for change | For logistical reasons the sexual hormones were measured both in male and female. After technical adaptations have been implemented – it is possible to perform the sexual hormone measurements in male subjects only. |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11.4 GLOBAL AMENDMENT 4

| Date of amendment | 20 Apr 2022 | |
|---|---|---|
| EudraCT number | 2021-004880-28 | |
| EU number | 2021 004000 20 | |
| BI Trial number | 1402-0020 | |
| BI Investigational Medicinal | BI 1358894 | |
| Product(s) | 21 100000 | |
| Title of protocol | Relative bioavailability of two different tablet | |
| Time of protocol | formulations of BI 1358894 administered in he | ealthy |
| | subjects in fasted and fed state (an open-label, | |
| | randomised, single-dose, four-period, four-sequence | |
| | crossover study) | |
| | 1 2/ | |
| Substantial Global Amendmen | nt due to urgent safety reasons | |
| | The state of the s | |
| Substantial Global Amendmen | ıt | |
| Non-substantial Global Amendment | | |
| | | 1000 1000 |
| | | 100 |
| Section to be changed | 1. Flowchart | |
| | 2. Section 1.2.1 | |
| | | 3. Section 1.4.2 Risks. Table 1.4.2: 1 |
| | 4. Section 1.4.3 Discussion | |
| | 5. Section 3.3.2 Inclusion criteria | |
| | 6. Section 4.2.2.3 Contraception requirements | |
| | 7. Section 6.2.1 | |
| Description of change | | <ol> <li>Timepoints for counselling regarding</li> </ol> |
| | | contraception included + footnote 10 |
| | A CONTRACTOR OF THE PROPERTY O | Insertion of embryofetal development data |
| | 3. Insertion of teratogenic risk | |
| | 4. Adding benefit risk considerations | |
| | 5. Adaptation of contraceptive measures. | |
| | Double barrier method added for | |
| | - female participants with vasectomized | 1 |
| | partners. | |
| | | - female participants with tubal ligation |
| | | Details on possible barrier methods provided. |
| | 6. Adding counselling on contraception | |
| Dationals for shares | | 7. Adding counselling on contraception |
| Rationale for change | fetal development study with BI 1358894 | Recently available data from a pivotal embryo- fetal dayslapment study with BL1358804 in |
| | minipigs has shown a teratogenic potenti | The state of the s |
| | the compound detected at relevant human | |
| | the compound detected at relevant human | ш |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| doses. Since a teratogenic effect in humans cannot be excluded, pregnancy of trial participants must be avoided. 2. See 1) 3. See 1) 4. See 1) 5. See 1) |
|---|
| 6. See 1)<br>7. See 1) |



#### APPROVAL / SIGNATURE PAGE

Document Number: c36231686 Technical Version Number: 5.0

Document Name: clinical-trial-protocol-version-05

**Title:** Relative bioavailability of two different tablet formulations of BI 1358894 administered in healthy subjects in fasted and fed state (an open-label, randomised, single-dose, four-period, four-sequence crossover study)

#### Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Author-Trial Statistician | | 20 Apr 2022 13:06 CEST |
| Author-Clinical Trial Leader | | 20 Apr 2022 13:33 CEST |
| Approval-Clinical Program Leaders | | 20 Apr 2022 13:42 CEST |
| Verification-Paper Signature<br>Completion | | 20 Apr 2022 13:46 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c36231686Technical Version Number: 5.0

#### (Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|-------------|
|----------------------|-----------|-------------|